# 16.1.9 **Documentation of Statistical Methods**

Statistical Analysis Plan (Protocol No: AL-335-604) Version 1.0 dated 17-May-2017

# STATISTICAL ANALYSIS PLAN

# ALIOS BIOPHARMA

260 E. Grand Ave South San Francisco, CA 94080

A Phase 2a, Open-Label Study to Evaluate the Safety, Pharmacokinetics and Efficacy of the Combination of AL-335 and Odalasvir, with or without Simeprevir, in Treatment-Naïve Subjects with Genotype 1, 2 or 3 Chronic Hepatitis C infection with or without compensated Child Pugh A Cirrhosis

Protocol No: AL-335-604

SAP Version 1.0

SAP Date: 17 May 2017

# **Prepared by:**

inVentiv Health Clinical

This document contains confidential information of Nichi-Iko Pharmaceutical Co., Ltd. Any viewing or disclosure of such information that is not authorized in writing by Nichi-Iko Pharmaceutical Co., Ltd., is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.



CONFIDENTIAL

STATISTICAL ANALYSIS PLAN
ALIOS BIOPHARMA
AL-335-604
Page 2 of 75

# STATISTICAL ANALYSIS PLAN

### SIGNATURE PAGE

# **ALIOS BIOPHARMA**

260 E. Grand Ave South San Francisco, CA 94080

A Phase 2a, Open-Label Study to Evaluate the Safety,
Pharmacokinetics and Efficacy of the Combination of AL-335 and
Odalasvir, with or without Simeprevir, in Treatment-Naïve Subjects
with Genotype 1, 2 or 3 Chronic Hepatitis C infection with or without
compensated Child Pugh A Cirrhosis

Protocol No: AL-335-604

| as KAKUDA, Clinical Ph<br>S BIOPHARMA | armacologist | Approval Date |
|---|---|---|
| | | • May 18, 2017 |
| MCCLURE, Senior Medion S BIOPHARMA | cal Director | Approval Date |
| | | 18M 2017 |
| | | • 10 - 9 - 201) |
| DEMASI, Clinical Biosta<br>SEN R&D US | tistics Functional Leader | Approval Date |

Final 1.0: 2017-MAY-17

# TABLE OF CONTENTS

| 1. | | Introduction | 8 |
|---|---|---|---|
| 2. | | Study objectives | 8 |
| 2 | 2.1 | Primary objective | 8 |
| 2 | 2.2 | Secondary objectives | 8 |
| 3. | | Study methodology | 9 |
| 3 | 3.1 | Description of cohorts and groups (based on protocol version 8.1 of the 21st of Decc | ember 2016) 9 |
| 3 | 3.2 | Visit Windows and Phase Definitions | 10 |
| 4. | | Statistical considerations | 15 |
| 5. | | Description of study subjects | 17 |
| 5 | 5.1 | Definition of analysis sets | 17 |
| 5 | 5.2 | Subject disposition | 17 |
| 5 | 5.3 | Protocol deviations | 18 |
| 5 | 5.4 | Definition of subgroups | 18 |
| 6. | | Demographic data and baseline characteristics | 18 |
| $\epsilon$ | 5.1 | Demographic data | 18 |
| $\epsilon$ | 5.2 | Other baseline characteristics | 18 |
| $\epsilon$ | 5.3 | Medical and surgical history | 19 |
| $\epsilon$ | 5.4 | Previous and concomitant medications | 19 |
| $\epsilon$ | 5.5 | Compliance | 19 |
| 7. | | Pharmacokinetic data | 20 |
| 7 | 7.1 | Generalities | 20 |
| 7 | 7.2 | Plasma pharmacokinetic concentrations and parameters | 21 |
| | | 7.2.1 Plasma pharmacokinetic parameters | 21 |
| | | 7.2.2 Plasma pharmacokinetic analysis | 22 |
| 8. | | Safety data | 23 |
| 8 | 3.1 | Adverse events | 23 |
| 8 | 3.2 | Clinical laboratory data | 24 |
| 8 | 3.3 | Other safety parameters | 27 |
| | | 8.3.1 Vital signs data | 27 |
| | | 8.3.2 Electrocardiogram data | 28 |
| | | 8.3.3 Other safety parameters | 30 |
| 9. | | Efficacy data | 31 |
| 9 | 9.1 | Analysis Specifications | 31 |
| | | 0.1.1 Lavel of Cignificance | 21 |

| | 9.1.2 | Data Handling Rules | 31 |
|---|---|---|---|
| 9.2 | Prima | ry Efficacy Endpoint | 31 |
| | 9.2.1 | Definition | 31 |
| | 9.2.2 | Analysis Methods | 32 |
| 9.3 | Major | Secondary Endpoints | 32 |
| | 9.3.1 | Definitions | 32 |
| | 9.3.2 | Analysis Methods | 34 |
| 10. | Report | ing conventions | 34 |
| 11. | Appen | dices | 36 |
| 11.1 | App | pendix 1 - Schedule of assessments of the study | 36 |
| 11.2 | App | pendix 2 - Criteria for Potentially Clinically Significant Abnormalities (PCSA) | 44 |
| 11.3 | App | pendix 3 - List of tables, listings and figures included in the clinical study report | 45 |
| 11.4 | App | pendix 4: Events of special/clinical interest | 60 |
| | 11.4.1 | Search terms for Events of Special/Clinical Interest | 60 |
| | 11.4.2 | RASH – SMQ19.1 | 62 |
| | 11.4.3 | CARDIAC EVENTS - SMQ19.1 | 63 |

# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AE | Adverse Event |
| ATC | Anatomic Therapeutic Chemical |
| AUC | Area Under the Curve |
| $AUC_{0\text{-last}}$ | Area Under the Curve from time zero to last measurable plasma concentration |
| $\mathrm{AUC}_{0\text{-}	au}$ | Area Under the Curve during one dosing interval |
| $AUC_{0\text{-}inf}$ | Area Under the Curve from time zero to infinity |
| BLQ | Below the Limit of Quantification |
| BMI | Body Mass Index |
| $C_{last}$ | Last measurable plasma concentration |
| $C_{\text{max}}$ | Maximum observed plasma concentration |
| $C_{\text{min}}$ | Minimum observed plasma concentration |
| CI | Confidence Interval |
| CL/F | Apparent oral clearance |
| CRF | Case Report Form |
| CV | Coefficient of Variation |
| ECG | ElectroCardioGram |
| i.e. | id est |
| HCV | Hepatitis C Virus |
| ICH | International Conference on Harmonization |
| IMP | Investigational Medicinal Product (synonymous with "study drug") |
| IS | Included Set |
| $\lambda_z$ | Apparent terminal elimination rate constant |
| LLN | Lower Limit of Normal range |

| Abbreviation | Definition |
|---|---|
| MedDRA <sup>®</sup> | Medical Dictionary for Regulatory Activities® |
| NCA | Non-Compartmental Analysis |
| PCSA | Potentially Clinically Significant Abnormalities |
| PK | PharmacoKinetics |
| PKS | PharmacoKinetic Set |
| PPS | Per Protocol Set |
| PT | Preferred Term |
| QRS | QRS interval duration |
| QT | Time interval for ventricular depolarisation and repolarisation |
| QTc | Corrected QT interval |
| QTcB | Bazett corrected QT interval |
| QTcF | Fridericia corrected QT interval |
| RAV | Resistance-Associated Variants |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| $\mathrm{SAS}^{\scriptscriptstyle{\circledR}}$ | Statistical Analysis System® |
| SD | Standard Deviation |
| SEM | Standard Error of the Mean |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| SVR | Sustained Virologic Response |
| t <sub>1/2</sub> | Apparent terminal elimination half-life |
| TFLs | Tables, Figures, and Listings |
| $t_{last}$ | Time corresponding to last measurable plasma concentration |
| $t_{max}$ | Time to reach maximum plasma concentration |

| Abbreviation | Definition |
|--------------|----------------------------------|
| TEAE | Treatment Emergent Adverse Event |
| ULN | Upper Limit of Normal range |
| VL | Viral load |
| Vz/F | Apparent volume of distribution |
| WBC | White Blood Cell |
| WHO | World Health Organisation |

### 1. Introduction

The Statistical Analysis Plan (SAP) details the statistical methodology to be used in analyzing study data and outlines the statistical programming specifications, tables, figures and listings. It applies to the whole study on final analysis. Viral sequencing (e.g., Resistance-Associated Variants (RAV)) analyses will be described in a separate SAP.

# 2. Study objectives

# 2.1 Primary objective

The primary objective of this study is as follows:

 To evaluate the safety and tolerability of AL-335 in combination with ODV with or without SMV in subjects with GT1 or GT2 or GT3 CHC infection in treatment-naïve subjects with or without compensated Child Pugh A Cirrhosis

#### 2.2 Secondary objectives

The secondary objectives of this study are as follows:

- To evaluate the efficacy of treatment with AL-335 in combination with ODV±SMV in subjects with GT1 or GT2 or GT3 CHC infection
- To evaluate the pharmacokinetics of AL-335 (and metabolites), ODV±SMV in plasma
- To evaluate the dynamics of HCV RNA in subjects with GT1 or GT2 or GT3 CHC infection treated with AL-335 in combination with ODV±SMV
- To evaluate the effect of baseline host and disease-related characteristics on treatment outcome
- To evaluate the impact of the presence of an (NS) 3 polymorphism (e.g., Q80K; SMV-containing arms only) and/or NS5A and NS5B polymorphisms at baseline on treatment outcome
- To evaluate the viral resistance profile after ≤12 weeks administration of AL-335 in combination with ODV±SMV

# 3. Study methodology

# $3.1\;$ Description of cohorts and groups (based on protocol version 8.1 of the 21st of December 2016)

| Cohort<br># | GТ | Cirrhosis | AL-335 dose<br>(mg) | ODV dose<br>(mg) | SMV dose<br>(mg) | Duration<br>(weeks) |
|---|---|---|---|---|---|---|
| 1 | 1 | N | 400 | 50 QD | 100 | 8 |
| 1b | 1 | N | 800 | 50 QOD | - | 8 |
| 2 | 1 | N | 800 | 50 QOD | 75 | 8 |
| 3 | 1 | N | 800 | 50 QOD | 75 | 6 |
| 4 | 1 | N | 800 | 50 QOD | | 8 (N=5)<br>12 (N=8) |
| 5 | 3 | N | 800 | 50 QOD | 75 | 8 (N=5)<br>12 (N=14) |
| 6 | 1 | Y | 800 | 50 QOD | 75 | 8 |
| 7 | 1 | Υ | 800 | 25 QD | 75 | 8 |
| 8 | 1 | Υ | 800 | 25 QD | 75 | 8 |
| 9 | 1 | Υ | 800 | 25 QD | 75 | 12 |
| 10 | 1 | Υ | 800 | 25 QD | 75 | 12 |
| 11 | 2 | Υ | 800 | 25 QD | 75 | 12 |
| 12 | 2 | Υ | 800 | 25 QD | 75 | 8 |
| 13-15 | TBD | | | | | |

| Cohort # | Genotype | Cirrhosis | AL-335<br>dose (mg) | ODV<br>dose (mg) | SMV<br>dose (mg) | Duration (weeks) | Group* |
|---|---|---|---|---|---|---|---|
| 1 | 1 | No | 400 | 50 QD | 100 | 8 | 1 |
| 1b | 1 | No | 800 | 50 QOD | - | 8 | 1b+4 |
| 2 | 1 | No | 800 | 50 QOD | 75 | 8 | 2 |
| 3 | 1 | No | 800 | 50 QOD | 75 | 6 | 3 |
| 4 | 1 | No | 800 | 50 QOD | - | 8 (N=5) | 1b+4 |
| | | | | | | 12 (N=8) | |

| 5 | 3 | No | 800 | 50 QOD | 75 | 8 (N=5)<br>12 (N=14) | 5 |
|---|---|---|---|---|---|---|---|
| 6 | 1 | Yes | 800 | 50 QOD | 75 | 8 | 6+7+8 |
| 7 | 1 | Yes | 800 | 25 QD | 75 | 8 | 6+7+8 |
| 8 | 1 | Yes | 800 | 25 QD | 75 | 8 | 6+7+8 |
| 9 | 1 | Yes | 800 | 25 QD | 75 | 12 | 9+10 |
| 10 | 1 | Yes | 800 | 25 QD | 75 | 12 | 9+10 |
| 11 | 2 | Yes | 800 | 25 QD | 75 | 12 | 11 |
| 12 | 2 | Yes | 800 | 25 QD | 75 | 8 | 12 |
| 13-15 | To be dete | To be determined | | | | | |

<sup>\*</sup>These are combined groups for presentation purpose of all data except pharmacokinetics,

# 3.2 Visit Windows and Phase Definitions

Phases will be constructed as follows:

| Trial phase | Start date | End date |
|---|---|---|
| Screening (phase 0) | Minimum of Date of signing the | 1 day before the first study drug intake (AL-335+ODV(±SMV)) |
| (P.1400 0) | informed consent and Date of the | |
| | first screening visit | |
| Treatment | Date of first study drug intake | Date of last study drug intake: |
| (phase 1) | (AL-335+ODV(±SMV)) | MAXIMUM{Date of last study drug intake (AL-335+ODV(±SMV))} + 3 days* |
| Follow-up | End date of Treatment phase | Trial termination date |
| (phase 2) | +1 | |

<sup>\*</sup>In case the last study drug intake is missing, other dates can be used instead for date of last study drug intake: E.g. if the subject discontinued treatment (known from the disposition table): date of the withdrawal visit, if the latter is not available: date of first available FU visit minus the number of days in follow-up at which this FU visit was scheduled according to the protocol. If those dates are not available, date of trial termination.

The number of days in the treatment phase (ADY) will be defined as:

 $ADY = visit\ date - date\ of\ first\ study\ drug\ intake\ +1$  for visits on or after the day of first study drug intake

 $ADY = visit\ date - date\ of\ first\ study\ drug\ intake$  for visits before the day of first study drug intake

In case the date of first study drug intake is missing, the date of the baseline visit can be used as date of first study drug.

Actual End of Treatment visit (EOT) is defined as the last visit in the Treatment phase.

All visits (regardless the investigated parameter) will be allocated within each phase to analysis time points based on the number of days in phase (ADY):

# **6-Week Cohorts**

| Trial phase | Target phase day | Analysis time point (numeric version) | Analysis time point <sup>b</sup> | Time<br>interval<br>(days) <sup>a</sup> |
|---|---|---|---|---|
| Screening | -∞ | -1 | Screening | <0 |
| | 1 | 0 | Baseline | ≤1 |
| | 2 | 0.2 | Day 2 | 2 |
| | 3 | 0.3 | Day 3 | [3,5] |
| | 7 | 1 | Week 1 | [6,11] |
| | 14 | 2 | Week 2 | [12,18] |
| | 21 | 3 | Week 3 | [19,25] |
| Treatment phase | 28 | 4 | Week 4 | [26,32] |
| | 35 | 5 | Week 5 | [33,39] |
| | 42 | 6 | Week 6 | [40, + ∞] |
| | last visit while on study therapy or 3 days after the day of last dose | 999 | ЕОТ | |
| Follow-up phase | 25 | 16 | Follow-up Week | [1,39] |

| 53 | 20 | Follow-up Week | [40,67] |
|-----|----|----------------------|-----------|
| 81 | 24 | Follow-up Week<br>12 | [68,102] |
| 123 | 30 | Follow-up Week | [103,144] |
| 165 | 36 | Follow-up Week 24 | [145, +∞] |

# 8-Week Cohorts

| Trial phase | Target phase day | Analysis time<br>point<br>(numeric<br>version) | Analysis time point <sup>b</sup> | Time<br>interval<br>(days) <sup>a</sup> |
|---|---|---|---|---|
| Screening | _∞ | -1 | Screening | <0 |
| | 1 | 0 | Baseline | ≤1 |
| | 2 | 0.2 | Day 2 | 2 |
| | 3 | 0.3 | Day 3 | [3,5] |
| | 7 | 1 | Week 1 | [6,11] |
| | 14 | 2 | Week 2 | [12,18] |
| | 21 | 3 | Week 3 | [19,25] |
| | 28 | 4 | Week 4 | [26,32] |
| Treatment phase | 35 | 5 | Week 5 | [33,39] |
| r | 42 | 6 | Week 6 | [40,46] |
| | 49 | 7 | Week 7 | [47,53] |
| | 56 | 8 | Week 8 | [54, +∞] |
| | last visit<br>while on<br>study therapy<br>or 3 days<br>after the day<br>of last dose | 999 | ЕОТ | |
| Follow-up phase | 25 | 16 | Follow-up Week 4 | [1,39] |
| | 53 | 20 | Follow-up Week 8 | [40,67] |
| | 81 | 24 | Follow-up Week 12 | [68,102] |
| | 123 | 30 | Follow-up Week | [103,144] |

| 165 | 36 | Follow-up Week | [145, +∞] |
|-----|----|----------------|-----------|
|-----|----|----------------|-----------|

# 12-Week Cohorts

| Trial phase | Target phase day | Analysis time<br>point<br>(numeric<br>version) | Analysis time point <sup>b</sup> | Time<br>interval<br>(days) <sup>a</sup> |
|---|---|---|---|---|
| Screening | _∞ | -1 | Screening | <0 |
| | 1 | 0 | Baseline | ≤1 |
| | 2 | 0.2 | Day 2 | 2 |
| | 3 | 0.3 | Day 3 | [3,5] |
| | 7 | 1 | Week 1 | [6,11] |
| | 14 | 2 | Week 2 | [12,18] |
| | 21 | 3 | Week 3 | [19,25] |
| | 28 | 4 | Week 4 | [26,32] |
| Treatment | 35 | 5 | Week 5 | [33,39] |
| phase | 42 | 6 | Week 6 | [40,46] |
| | 49 | 7 | Week 7 | [47,53] |
| | 56 | 8 | Week 8 | [54,60] |
| | 84 | 12 | Week 12 | [82, +∞] |
| | last visit<br>while on<br>study therapy<br>or 3 days<br>after the day<br>of last dose | 999 | ЕОТ | |
| Follow-up phase | 25 | 16 | Follow-up Week 4 | [1,39] |
| | 53 | 20 | Follow-up Week 8 | [40,67] |

| 81 | 24 | Follow-up Week | [68,102] |
|-----|----|-------------------|-----------|
| 123 | 30 | Follow-up Week | [103,144] |
| 165 | 36 | Follow-up Week 24 | [145, +∞] |

<sup>&</sup>lt;sup>a</sup> The reference day of the Treatment and Screening phase is the day of the first study drug intake (= day 1 in Treatment phase).

If two visits fall within the same interval, the last measurement within the interval will be used for the descriptive statistics/tabulations per time point and graphics in order to have only one evaluation per subject per analysis time point. If there are two measurements on the same day and time, then the measurement with the highest sequence number will be used. Listings will include all values.

### 4. Statistical considerations

Efficacy and safety data will be analysed using SAS® software version 9.4 (SAS institute Inc. USA).

Pharmacokinetic data from the PK substudy will be analysed using Phoenix<sup>®</sup> WinNonLin<sup>®</sup> version 6.4 (Pharsight) and SAS<sup>®</sup> software version 9.4 (SAS Institute Inc. USA) for final analysis.

Descriptive statistics will be supplied according to the nature of the criteria:

- Quantitative variable: sample size, arithmetic mean, standard deviation (SD), standard error of the mean (SEM), minimum, median and maximum, and quartiles if necessary (with geometric mean, arithmetic and geometric coefficients of variation (CV), and quartiles for PK parameters, geometric mean will not be reported in case of value equal to 0).
- Qualitative variable: sample size, absolute and relative frequencies per class. Percentages will be provided with one decimal place.

Safety data will be organized by cohort.

All safety and pharmacokinetics listings will be sorted by cohort, subject, and measurement time if applicable.

For all except pharmacokinetics data, cohorts that evaluate the same treatment regimen for the same duration (e.g., Cohort 1b and the first 5 subjects in Cohort 4) will be pooled (using Label "Cohort 1b+Cohort 4 (8 Weeks)." If multiple treatment durations and/or regimens were assessed in a single cohort, the data for that cohort will be presented separately (e.g. Cohort 4 (12 weeks) will be separate from Cohort 4 (8 weeks), which will be pooled with cohort 1b). For cohorts with different clinical characteristics (e.g. HCV genotype, cirrhosis status),

<sup>&</sup>lt;sup>b</sup> Target day in follow-up phase equals target day in the protocol minus 3 days.

treatment regimens or same treatment regimen but with different durations, data will be presented separately.

For pharmacokinetic data, cohorts that evaluate the same treatment regimen (including study medications and doses) in the same population (cirrhotic vs non-cirrhotic), whatever the duration, or HCV genotype will be pooled, i.e. the presentation of cohorts will be:

- Cohort 1,
- Cohort 1b+4,
- Cohort 2+Cohort 3+Cohort 5,
- Cohort 6.
- Cohort 7+Cohort 8+Cohort 9+Cohort 10+Cohort 11+Cohort 12

# Handling of missing and retest values

No management of missing data will be done, except for pharmacokinetic values (see section 7.1) and missing or incomplete start/stop dates (see below).

Missing start or end dates for events not aligned to a specific visit/week such as adverse events, medications reported, etc., will be imputed using the following rules:

- A completely missing start date of an event will be set to the date of the first dose of study medication, unless it is clearly indicated that this is an event happening pretreatment. In this case, it will be set to the day before the first dose of study medication.
- A completely missing stop date will not be imputed, but the event will be assumed to be ongoing.
- Partially missing dates where the year is known will be set to 01 January of that year
  or the first dose of study medication date, if the first dose of study medication
  occurred in that year.
- Partially missing dates where the year and month are known will be set to the first day
  of that month or the first dose of study medication date, if the first dose of study
  medication occurred in that month.

If, by applying the above rules, the stop date is imputed before the start date, then the stop date will be set to be the same as the start date.

For all parameters and for subjects with retest values, the last reliable value will be used as a measurement time before the first investigational medicinal product (IMP) administration (provided it was measured before IMP administration) and the first reliable value will be used as a measurement time after the first IMP administration.

#### **Baseline definition**

For all parameters, baseline will be defined as the last available (and reliable if applicable) single measurement prior to the first IMP administration unless otherwise specified (e.g. ECG).

### **Duration**

Duration (in days, hh:mm) will be calculated as the difference between start and stop date and time (e.g. duration of AE (days, hh:mm) = date of AE end date and time – date of AE onset date and time).

Duration (in days) will be calculated as the difference between start and stop date + 1 (e.g. duration of a medication (days) = date of medication end date - date of medication onset date + 1).

### Type I error rate

No significance testing will be performed. However, two-sided Clopper-Pearson 95% CI will be constructed around the proportion of subjects with sustained virologic response (SVRx) and other virologic response parameters, for each cohort.

# 5. Description of study subjects

#### 5.1 Definition of analysis sets

The following analysis sets will be defined:

Included set (IS): all the subjects included in the study.

<u>Safety/Efficacy/Intent-to-treat population (Safety set):</u> All subjects enrolled into the study who have received at least one dose of any study drug, whether prematurely withdrawn from the study or not, will be included in the safety/efficacy/Intent-to-treat set.

<u>Pharmacokinetic set (PKS): Will be comprised of all safety set</u> subjects except those that they significantly violate the inclusion or exclusion criteria, deviate significantly from the protocol or if data are unavailable or incomplete which may influence the PK analysis. Excluded cases will be documented together with the reason for exclusion.

<u>Per Protocol set (PPS)</u>: A per protocol analysis including all subjects enrolled and adherent to the protocol may be performed for certain efficacy analyses.

A subset of major protocol deviations, that may have an impact on the results of the analysis, will be identified prior to database lock. If there are a substantial number of subjects with such protocol deviations, a per-protocol analysis will be performed on the primary endpoint, based on subjects from the Safety set, excluding these subjects. Additional efficacy analysis using the PPS may be performed on an ad-hoc basis.

# 5.2 Subject disposition

A summary table with the description of the number of included subjects, the number of subjects who completed study and the number of subjects who discontinued classified by main reason of withdrawal will be performed by cohort and overall on the subjects included in the Included set. Corresponding individual listings will be provided.

A summary table with the description of the number and percentage of subjects in each analysis set (Safety set, and Pharmacokinetic set) will be performed by cohort and overall. A specific listing of subjects excluded from safety/efficacy and pharmacokinetic analyses will be provided with reason for exclusion.

A summary table with the number and percentage of subjects at each visit will be performed by cohort and overall on the subjects included in the safety set.

Listings with end of study status and study visit dates will also be carried out.

#### 5.3 Protocol deviations

A summary table by cohort and overall with the number and percentage of subjects presenting deviations relating to inclusion/exclusion criteria (all eligibility criteria responses) will be prepared on the subjects included in the safety set. A summary table by cohort and overall with the number and percentage of subjects presenting other protocol deviations (all deviations judged relevant by the sponsor during the data-review meeting) will also be prepared. The corresponding listings will be provided with the status of deviation (minor/major, as assessed by the sponsor during the data-review meeting).

### 5.4 Definition of subgroups

The following subgroups will be considered to be investigated for efficacy; combinations of more than one subgroup may also be done. In case subgroup categories are smaller than 10 subjects within a cohort, subgroup categories might be combined.

- IL28B genotype (CC, CT, TT)
- HCV genotype/subtype (1a,1b, 1other, 2, 3)
- Prior treatment status (cirrhosis cohorts only) prior pegylated interferon + ribavirin treatment with relapse

# 6. Demographic data and baseline characteristics

The analyses on demographic and other baseline characteristics will be performed on the safety set and PK set. Analyses on medical and surgical history, previous and concomitant medication, and compliance will be performed for the safety set.

Separate ad hoc summary tables of the demographic data and baseline characteristics for all subjects in cohorts 1b+4 (N=33) and cohort 5 (N=19) will be generated since, at the time of enrolment, all subjects in these two groupings were intended to dose for the same duration.

#### 6.1 Demographic data

Subjects' demographic characteristics (age, sex, race, ethnicity, height, weight and BMI recorded at screening and Interleukin 28B genotype) will be summarised by cohort and overall, and listed.

#### 6.2 Other baseline characteristics

HCV genotype as well as HCV RNA values at baseline (in IU/mL and log<sub>10</sub> IU/mL) will be summarised by cohort and overall, and listed.

Serology testing will be listed.

Positive results of serology will be listed.

Childbearing status (for female only) and contraception method will be listed.

Alcohol consumption will be listed.

Information related to liver biopsy and fibroscan will be listed as well as Child-Pugh class assessment and hepatocellular carcinoma assessment (only for compensated cirrhosis cohort). Fibroscan score and Child-Pugh score will be summarised by cohort and overall.

# 6.3 Medical and surgical history

Information on medical and surgical history recorded at the screening visit will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA®) Version 19.1.

A table with the number and percentage of subjects having at least one previous/ongoing medical and surgical history (except liver diseases) will be generated by cohort and overall. The same table will be provided for liver diseases (SOC: "Hepatobiliary disorders"). Previous/ongoing medical and surgical history (except liver diseases) and previous/ongoing medical and surgical history related to liver diseases will be listed separately.

### 6.4 Previous and concomitant medications

Information on previous and concomitant medications will be coded according to the WHO drug Dictionary (WHO-DD) version of June 2015.

A previous medication will be defined as a medication stopped prior to the date and time of first administration of IMP. A concomitant medication will be defined as a medication which is taken by subjects any time during the treatment period (on or after the date and time of first IMP administration for each subject).

Incomplete dates (i.e. day and/or month and/or year missing):

- In case of a partial start date, the therapies are allocated to the phases using the available partial information, no imputation is done. If, for instance, for a therapy start date only month and year is available, these data are compared with the month and year info of the phases.
- In case of a completely missing start date, the therapy is considered as having started before the trial. In case of a completely missing end date, the therapy is considered as ongoing at the end of the trial.
- In case of a partial end date, the therapies are allocated to the phases using the available partial information, no imputation is done. If, for instance, for a therapy end date only month and year is available and are the same as month and year of the first IMP administration, the therapy is considered as concomitant.

A table with the number and percentage of subjects having at least one previous medication will be generated by cohort and overall (overall and by Anatomical Therapeutic Chemical (ATC) and by preferred name). A table with the number and percentage of subjects having taken at least one concomitant medication will be generated by cohort and overall (overall and by Anatomical Therapeutic Chemical (ATC) and by preferred name). Previous and concomitant medications will be listed separately.

### 6.5 Compliance

A listing with IMP administration dates and times will be carried out for each study drug. Subjects that took additional doses (either extra doses on a dosing day (all drugs) or on

additional days other than those planned (for ODV QOD regimens) will be flagged in the listing. Time of meals intake will be listed as well.

#### 7. Pharmacokinetic data

Two types of PK analysis will be performed for this study: 1) Non-compartmental analysis (NCA) for subjects participating in the PK substudy and 2) population PK in all subjects. This SAP will only cover the NCA PK analyses done in patients in the PK substudy. The population PK analysis will be described in a separate SAP and will have its own report.

The pharmacokinetic analysis will be performed on the pharmacokinetic set (PKS).

#### 7.1 Generalities

The following rules for **PK parameters calculation** after each administration will be used:

Actual sampling times will be used for deriving PK parameters. In the case the actual sampling time will not be known, the scheduled time will be used, with appropriate footnoting. Actual sampling times will be checked for major aberrations. In case a major aberration occurs for an actual sampling time (i.e., >20.00% deviation from the scheduled time), this plasma concentration will be excluded from descriptive statistics in the plasma concentration table and reported in the CSR.

If an entire concentration-time profile is below the limit of quantification (BLQ), the profile will be excluded from the PK analysis.

All BLQ values will be replaced by "0".

All embedded BLQ values (BLQ value between two measurable concentrations) will be treated as missing. Details of this exclusion must be documented in the clinical study report.

For the determination of  $\lambda_z$ , only those data points judged to describe the terminal log-linear decline resulting in an adjusted coefficient of determination value > 0.9 will be used in the regression. A minimum of 3 data points will be used in calculating  $\lambda_z$  (excluding  $C_{max}$ ). The number of points and the lower and upper limits of the terminal phase will be identified in the study data and in the CSR.

If there are late positive concentration values following 2 BLQ concentration values in the apparent terminal phase, these values will be evaluated. If these values are considered to be anomalous or to introduce a substantial bias, they will be set to missing and excluded from the PK analysis.

The following rules for **plasma concentration versus time graphic representation** will be used:

No graphic representation will be made if all values are BLQ.

All BLQ values will be replaced by "0".

All BLO values will not be shown on semi-logarithmic plots.

Profiles and individuals values considered to be outliers should be included in the individual plots and excluded in the mean plots.

Actual sampling times will be used for individual subjects PK profiles and nominal sampling times should be used for mean plots.

All subjects will be plotted with the same scale and range of values on the x- and y-axes

The following rules for mean plasma concentration calculation will be used:

If more than half (>50%) of the values at a single time point are BQL, mean and median values will be reported as BQL. Standard deviation and %CV will not be reported; maximum and minimum values will be reported as observed (including BQL).

If more than (or equal) half of values are not BLQ: statistics will be calculated considering BLQ values as zero.

# For summary statistics for PK parameters:

If more than (or equal to) half of values are available: statistics will be calculated considering available values.

If less than half of values are present: mean will not be calculated and presented as missing. Min, median and max value on available values will be presented.

All concentrations below the limit of quantification or missing data will be labelled as such in the concentration data listings.

# 7.2 Plasma pharmacokinetic concentrations and parameters

# 7.2.1 Plasma pharmacokinetic parameters

Blood samples will be drawn for AL-335, SMV and ODV (depending on the cohorts) on:

- On Day 1 at 0 hour,
- On Week 2 at 0, 0.5, 1, 2, 3, 4, 6, 9, 12 and 24 hours (For PK substudy only),
- On Week 3 at 0, 2-4 hours,
- On Week 4 at 0, 6-8 hours,
- On Week 6 at 0, 2-4 hours,
- On Week 8 at 0, 6-8 hours (8 or 12 Week Cohorts),
- On Week 10 at 0, 2-4 hours (12 Week Cohorts),
- On Week 12 at 0, 6-8 hours (12 Week Cohorts).

For subjects in the PK substudy, relevant plasma pharmacokinetic (PK) parameters will be calculated for AL-335 and its metabolites (ALS-022399 and ALS-022227), SMV and ODV by standard non-compartmental methods for those subjects with sufficient plasma concentration data. The rules defined in the previous section 7.1 will be used.

The different areas under the concentration-time curve (AUC) will be calculated using the linear Trapezoidal summation (both ascending and descending phase).

The following plasma pharmacokinetic parameters will be calculated for AL-335 and its metabolites (ALS-022399 and ALS-022227), SMV and ODV:

| Parameters (unit) | Definition |
|---|---|
| C <sub>min</sub> (unit) | Minimum observed plasma concentration |
| C <sub>max</sub> (unit) | Maximum observed plasma concentration |
| C <sub>trough</sub> (unit) | Concentration at the end of a dosing interval before the next dose administration (Pre-dose or $C_{0h}$ ) |
| $t_{max}(h)$ | Time to reach maximum plasma concentration |
| AUC <sub>0-last</sub> (unit.h) | Area under the plasma concentration-time curve from time zero to last measurable (Non-BLQ) plasma concentration |
| | In cases where a subject's $AUC_{0-last}$ is estimated over a time interval that is very different from that of the other subjects in the group, it is recommended that subject's $AUC_{0-last}$ could be excluded from the calculation of descriptive statistics. All exclusions must be clearly documented in the CSR. |
| | In cases where more than half of subjects have a different $t_{last}$ , it may not be appropriate for the descriptive statistics for $AUC_{0-last}$ to be reported. |
| AUC <sub>0-24</sub> (unit.h) | Area under the plasma concentration-time curve from time zero to 24 hours |
| AUC <sub>0-48</sub> (unit.h) | Area under the plasma concentration-time curve from time zero to 48 hours (only for ODV and QOD cohorts) |
| $C_{ss,avg}$ | Average concentration of the drug calculated as follows: |
| | $C_{ss,avg} = AUC_{0-\tau} / \tau$ |
| C <sub>last</sub> (unit) | Last observed plasma concentration |
| t <sub>last</sub> (h) | Time to reach last plasma concentration |

# 7.2.2 Plasma pharmacokinetic analysis

Listings with plasma concentrations of AL-335, ALS-022399 and ALS-022227, SMV and ODV (including PK blood sampling dates and times) and PK parameters will be provided by cohort, dose, and subject. These listings will be performed on all subjects with an available profile (complete or incomplete), including those who are excluded from the PKS.

A specific listing will be also done focussing on subjects who either discontinue the study for an adverse event, experience a severe adverse event or a serious adverse event.

Individual plasma concentrations for all subjects and PK parameters of AL-335, ALS-022399 and ALS-022227, SMV and ODV including descriptive statistics for subjects participating in the PK substudy will be presented in tables by cohort and by pooled cohorts.

Graphs for plasma concentration versus time profiles of AL-335, ALS-022399 and ALS-022227, SMV and ODV will be generated on linear and log/linear coordinates for arithmetic mean (±SD) by cohorts.

In addition, the plasma concentration versus time profiles of AL-335, ALS-022399 and ALS-022227 will also be presented on the same graph or as a separate graph on linear and log/linear coordinates for arithmetic mean (±SD) by pooled cohort.

Moreover, the plasma concentration versus time profiles of AL-335, ALS-022399 and ALS-022227, SMV and ACH-3102 will be presented graphically on linear and log/linear coordinates for each subject.

Pre-dose ("trough") concentrations of AL-335, ALS-022399 and ALS-022227, SMV and ODV for all subjects at all available timepoints will be presented graphically on linear coordinates for arithmetic mean (±SD) by cohorts and by pooled cohorts.

Scatter plots will be generated for the comparison of  $C_{trough}$ ,  $C_{max}$ , and  $AUC_{0-\tau}$  parameters of AL-335, ALS-022399, ALS-022227, SMV and ODV by cohorts and by pooled cohorts.

# 8. Safety data

The safety analyses will be performed on the safety set.

#### 8.1 Adverse events

Adverse events, including pre-treatment events, will be recorded from the time of consent through the completion visits, for the treatment and follow-up phase combined.

Adverse events will be coded according to MedDRA® Version 19.1.

A treatment-emergent adverse event (TEAE) is an adverse event that occurs after the first IMP administration or that was present prior to dosing but exacerbated after the first IMP administration.

Adverse events will be summarised in tables as follows (overall and by System Organ Class (SOC) and Preferred Term (PT)):

- Number and percentage of subjects with at least one adverse event and number of adverse events for each cohort,
- Number and percentage of subjects with at least one TEAE and number of TEAEs for each cohort,
- By intensity, with the number and percentage of subjects with at least one TEAE and number of TEAEs for each cohort,
- By causality of each treatment, with the number and percentage of subjects with at least one TEAE and number of TEAEs for each cohort.

Moreover, an overall summary table of all TEAEs will be presented.

In addition, summary tables will also be presented for TEAEs, serious TEAEs, TEAEs leading to any study drug discontinuation, severe or life threatening (i.e. Grade 3 / 4) TEAEs, and TEAEs with fatal outcome by decreasing frequency of PT.

The incidence and comparable prevalence rate per 2-week time interval for any AEs will be summarized and plotted by cohort.

Note: Repetitions will only be counted once in summary tables. Repetitions are defined as follows: if a given subject presents several adverse events with the same preferred term during the same phase (treatment and follow-up phase combined), only one event is counted, the others are considered repetitions or recurring episodes. The start time of the event will be the start time of the first occurrence, the end time will be the end time of the last episode. The intensity will be the highest recorded intensity for all episodes. The causality will be the highest likelihood recorded for all episodes.

A summary table of TEAEs of special interest (cardiac events, increased bilirubin (hyperbilirubinemia, blood bilirubin increased), rash and photosensitivity) will be also presented (see Appendix 4 for detailed list of SMQs).

The incidence rates for each event of interest by WHO toxicity grades and relationship to study drugs will be summarized. Time to the first occurrence of the events of interest will be summarized and Kaplan-Meier curves will be plotted.

The incidence and comparable prevalence rate per 2-week time interval for AEs of special interest will be summarized and plotted by cohort.

Bar graphs of the worst toxicity grade of cardiac events over time by cohort will be plotted.

All adverse events for subjects who met the Study Stopping Rules(i.e. <1 log decline in HCV RNA after 4 weeks of treatment) will be listed.

All TEAEs reported in the CRF will be listed with the SOC, PT and investigator's verbatim. Additional listings will be provided for serious adverse events (SAEs), TEAEs with grade 3 or grade 4, TEAEs leading to any study drug discontinuation, TEAEs of special interest, and TEAEs with fatal outcome.

In case of rash, all information related to rash assessments will be listed.

#### 8.2 Clinical laboratory data

The following clinical laboratory parameters will be measured (see section 12.1):

- At the screening visit,
- On Day 1, Week 1, Week 2, Week 4, Week 6, Week 8 (8 or 12 Week Cohorts), Week 10 (12 Week Cohorts), Week 12 (12 Week Cohorts), safety follow-up visit.

Additional measurements are done on Week 3, Week 5 and Week 7 for alanine aminotransferase (ALT) and aspartate aminotransferase.

**Haematology** parameters will be listed and grouped as follows:

- Red blood cells: haemoglobin (g/L), haemoglobin A1C (mmol/mol) only at screening, hematocrit (fraction of 1), mean corpuscular haemoglobin (MCH) (fmol), mean corpuscular

haemoglobin concentration (MCHC) (mmol/L), mean corpuscular volume (MCV) (fL), mean platelet volume (MPV) (fl), erythrocyte sedimentation rate (mm/h), red distribution width (RDW) (%), reticulocytes (G/L and %) and red blood cell count (RBC) (T/L).

- White blood cells: basophils (G/L and %), eosinophils (G/L and %), lymphocytes (G/L and %), monocytes (G/L and %), neutrophils (G/L and %)) and white blood cell count (WBC) (G/L).
- Platelets (G/L).

# **Blood chemistry parameters** will be listed and grouped as follows:

- <u>Liver function</u>: alanine aminotransferase (ALT) (IU/L), alkaline phosphatase (IU/L), aspartate aminotransferase (AST) (IU/L), total bilirubin ( $\mu$ mol/L) and direct bilirubin ( $\mu$ mol/L).
- Renal chemistry: creatinine (µmol/L) and blood urea nitrogen (BUN) (mmol/L).
- <u>Electrolytes</u>: calcium (mmol/L), chloride (mmol/L), phosphorus (mmol/L), potassium (mmol/L), sodium (mmol/L) and bicarbonates (mmol/L).
- <u>Metabolism parameters</u>: glucose (mmol/L), cholesterol (mmol/L), triglycerides (mmol/L), lipase (IU/L), uric acid (µmol/L) and lactate dehydrogenase (LDH) (IU/L).
- Other parameters: albumin (g/L), creatine kinase (CPK) (IU/L), total protein (g/L), alpha fetoprotein (ug/L) only at screening, Alpha-1 Acid Glycoprotein (g/L) only at screening, Beta natriuretic peptide (BNP) and NT-pro-BNP.

# Coagulation parameters will be listed and grouped as follows:

- <u>Coagulation parameters</u>: prothrombin time (PT) (s), activated partial thromboplastin time (aPTT) (s) and international normalized ratio (INR).

**Urinalysis** parameters will be listed and grouped as follows:

- <u>Planned urinalysis parameters</u>: dipstick determination of pH, specific gravity, glucose, bilirubin, ketones, leukocytes, nitrite, occult blood, protein and urobilinogen.
- <u>Direct microscopy</u>: in case of abnormal urinalysis parameters (in listing only).

Hormonology parameters will be listed as follows: FSH (IU/L) and estradiol (pmol/L)

In case a laboratory test result is *censored* (no numeric value is available, but only a verbatim term), the following rules are applied:

- < x or > x → a numeric value will be imputed by a value exceeding the cut-off value with one unit.
- $\leq x \text{ or } \geq x \Rightarrow \text{ imputation by } x.$

Laboratory values will be graded based on the following toxicity grading scale: The Division of AIDS Table for Grading the Severity of Adult and Pediatric AEs ("DAIDS grading table", version of November 2014), Appendix F - protocol version 8.0 of the 13<sup>rd</sup> of September 2016.

Lab values will also be graded based on WHO grading scale, but summary tables will be based on DAIDS grading scale only.

For haematology, blood chemistry, and coagulation, raw data and changes from baseline (Day 1) if applicable will be described by measurement time, for each cohort.

For all lab parameters with toxicity grade, a summary table with the number and percentage of subjects with treatment emergent grade 1-4 and 3+4 will be generated for each cohort for the worst post-baseline value. The same table will be provided by measurement time.

For haematology and blood chemistry, graphs of individual subject values (spaghetti plots) will be generated for each cohort for the following parameters: ALT, AST, alkaline phosphatase, total bilirubin, direct bilirubin, blood urea nitrogen, creatinine, CPK, BNP, haemoglobin, platelets and white blood cells.

A listing of all values of a parameter over time for any parameter with treatment emergent Grade 3 or 4 will be generated. A listing of all values of a parameter over time for any parameter with treatment emergent abnormal values will be also generated.

Values will be listed (raw data and change from baseline) and laboratory abnormal values will be flagged with their toxicity grades and clinical significance information.

For urinalysis, raw data will be described by measurement time, for each cohort.

Urinalysis values will be listed including direct microscopy if any.

Hormonology parameters will be listed only.

For applicable lab parameters, cross-tabulation of the worst toxicity grades versus baseline will be presented, Plots of mean(SE), mean(SE) of change from baseline by cohort over time and Bar graphs of the treatment emergent abnormality by toxicity grade over time for selected laboratory parameters will be plotted.

In determining DAIDS toxicity grades the following rules are applied:

- The worst grades/abnormalities are determined over the whole observational period, including all post-reference scheduled and unscheduled measurements.
- The abnormalities "abnormally low" and "abnormally high" are considered equally important, i.e. if a subject has an "abnormally low" as well as an "abnormally high" post-reference value, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%)
- If, for a specific test, the grading list provides distinct limits for abnormally low (=hypo) values as well as for abnormally high (=hyper) values, this test should be repeated for hyper and hypo limits separately in cross-tabulations and in the ADaM database.

For the grades, no distinction will be made between test results of samples obtained under fasting and under non-fasting conditions: in case limits under fasting and non-fasting conditions differ, the limits of the conditions (fasting/non-fasting) of scheduled visits as planned in the CTP will always be used, also for samples obtained under a different condition (e.g. samples of withdrawal visits).

Definition treatment-emergent: An abnormality (toxicity grade or abnormality based on normal ranges) will be considered treatment-emergent in a particular phase if it is worse than the reference. If the reference is missing, the abnormality is always considered as treatment-emergent. A shift from "abnormally low" at reference to "abnormally high" post reference (or vice versa) is also treatment-emergent.

#### 8.3 Other safety parameters

# 8.3.1 Vital signs data

Blood pressures (diastolic [DBP] and systolic [SBP]; mmHg), respiratory rate (breaths/min), body temperature (°C) and pulse rate (bpm) will be measured (see section 12.1) for each cohort at the screening visit, Day 1, Week 1 and then once a week thereafter.

Raw data and changes from baseline (Day 1 pre-dose) will be described by measurement time, for each cohort.

A summary table with the number and percentage of subjects with PCSA values (defined in section 12.2) will be generated by measurement time, for each cohort.

A specific listing of all values of a parameter over time for any parameter with PCSA values with clinical significance information will be generated.

| Pulse rate, DBP | , and SBP | are classified | in the fol | lowing a | bnormality c | odes: |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

| | Pulse (bpm) | DBP (mmHg) | SBP (mmHg) |
|---------------------|-------------|---------------|---------------|
| Abnormally low | ≤ 50 | ≤ 50 | ≤ 90 |
| Abnormally high | ≥ 120 | - | - |
| Grade 1 or mild | - | > 90 - < 100 | > 140 - < 160 |
| Grade 2 or moderate | - | ≥ 100 - < 110 | ≥ 160 - < 180 |
| Grade 3 or severe | - | ≥ 110 | ≥ 180 |

A summary table with the number and percentage of subjects with abnormal values (as defined above) will be generated for each cohort for the worst post-baseline value. The same table will be provided by measurement time.

A specific listing of all values of a parameter over time for any parameter with abnormal values with clinical significance information will be generated.

Values (raw data and changes from baseline) will be listed and PCSA and abnormal values will be flagged with clinical significance information.

Graph of mean (SE) by cohort over time will be plotted.

In determining the abnormalities, the following rules are applied:

 Worst grades/abnormalities are determined over the whole observational period, including post-baseline scheduled and unscheduled measurements. - The abnormalities 'abnormally low' and 'abnormally high'/grades are considered equally important, i.e. if a subject has an 'abnormally low' as well as an 'abnormally high' or graded post-baseline value, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%.)

# Definition treatment-emergent:

An abnormality will be considered treatment-emergent if it is worse than the baseline. If the baseline is missing, the abnormality is always considered as treatment-emergent. A shift from 'abnormally low' at baseline to 'abnormally high' or 'grade 1' or 'grade 2' or 'grade 3' post baseline (or vice versa) is also treatment-emergent.

### 8.3.2 Electrocardiogram data

Standard 12-lead ECG parameters (including heart rate (bpm), PR interval (ms), QRS duration (ms), QT interval (ms), Bazett QTc interval (QTcB; ms) and Fridericia QTc interval (QTcF; ms)) from both automatic and centrally read data, information on T- (normal or abnormal) and U-waves (normal or abnormal) and ECG abnormality will be measured (see section 12.1) for each cohort at the screening visit, Day 1, Week 1 and then once a week thereafter.

The mean of the triplicate ECGs will serve as analysable data for each visit. If one or more assessment is missing/not done then the mean will be calculated using the available assessments.

Centrally read data will be used for summary statistics and both locally and centrally read data will be listed.

Raw data and changes from baseline (Day 1 pre-dose) (except for T-and U-wave and ECG abnormality) will be described by measurement time, for each cohort.

A summary table with the number and percentage of subjects with PCSA values (defined in section 12.2) will be generated by measurement time, for each cohort.

Graphs of individual subject values (spaghetti plots) will be generated for each cohort for the following parameters: PR, QRS, QTcB, and QTcF. These graphs will include indications for the most conservative upper and lower limit of normal.

A specific listing of all values of a parameter over time for any parameter with PCSA values with clinical significance information will be generated.

A listing of all values over time for subjects with any clinically significantly abnormal ECGs will also be generated.

A listing of subjects with potentially progressive PR prolongation will be generated.

Potentially progressive PR prolongation is defined as any subject who has a post-baseline change of >20 ms from the highest pre-dose value.

Values (raw data/T- and U-wave/ECG abnormalities and changes from baseline) will be listed and data out of PCSA range will be flagged with clinical significance information.

The following abnormality categories are defined:

| | ECG parameter | | | |
|---|---|---|---|---|
| Abnormality Code | HR | PR | QRS | QT <sub>corrected</sub> * |
| Abnormalities on actual values | | | | |
| Abnormally low | ≤50 bpm | <120 ms | NA | = |
| | ≥120 bpm | ]200-240] ms | >120 ms | = |
| Abnormally high | | ]240-300] ms | | |
| | | >300 ms | | |
| Borderline: ]450 ms, 480 ms] | - | - | - | 450 ms< QTc ≤480 ms |
| Prolonged: ]480 ms, 500 ms] | - | - | - | 480 ms< QTc ≤500 ms |
| Pathologically prolonged: >500 ms | - | - | - | QTc>500 ms |
| Abnormalities on increase from | | | | |
| baseline | | | | |
| | - | [30; 60] ms | - | [30; 60] ms |
| | - | >60 ms | - | >60 ms |

<sup>\*</sup> QTcB or QTcF

A summary table with the number and percentage of subjects with abnormal values (as defined above) will be generated for each cohort for the worst post-baseline value. The same table will be provided by measurement time.

A specific listing of all values of a parameter over time for any parameter with abnormal values with clinical significance information will be generated.

A specific listing of all overall interpretations over time for any subject with any overall interpretation considered to be clinically significantly abnormal will be created.

In determining the abnormalities, the following rules are applied:

- Worst abnormalities are determined over the whole observational period, including post-baseline scheduled and unscheduled measurements.
- The abnormalities 'abnormally low' and 'abnormally high' are considered equally important, i.e. if a subject has as well an abnormally low as an abnormally high post-baseline, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%).

Cross-Tabulation of the worst ECG abnormalities in actual value versus the baseline value and Cross-Tabulation of the worst QTc increase versus the abnormality on the actual value will be presented.

Graphs of actual mean(SE), mean of change from baseline(SE) by cohort over time will be plotted. Spaghetti plots of PR for the patients who had prolonged PR interval or AV block (grade>=1) will be plotted.

# Definition treatment-emergent:

An abnormality will be considered treatment-emergent if it is worse than the baseline. If the baseline is missing, the abnormality is always considered as treatment-emergent. A shift from 'abnormally low' at baseline to 'abnormally high' or 'grade 1' or 'grade 2' or 'grade 3' post baseline (or vice versa) is also treatment-emergent.

### 8.3.3 Other safety parameters

Echocardiograms will be performed at regular intervals and according to a standard protocol.

The centrally read echocardiogram results will be used for analysis.

The maximum decline in mean ejection fraction (EF) from baseline will be summarized in a table by cohort with the following cutoffs: decline of >10%, decline of >5- $\le$ 10% and decline of >0-<=5%. Moreover, the number of subjects with any mean EF that declines by >10%, >5- $\le$ 10% or >0-<=5% will be summarized by measurement time and cohort.

A listing of all mean EFs by time point for subjects with any mean EF that declines by >10% or  $>5-\le10\%$  will be provided.

Moreover, for the following parameters: diastolic volume, left ventricular ejection fraction (LVEF) single plane, LV fractional shortening, LVPW diastolic thickness, systolic volume and ventricular septum diastolic thickness, the following analyses will be performed:

Raw data and changes from baseline (Screening) as well as percent changes from baseline will be described by measurement time, for each cohort.

Graphs of individual subject values (spaghetti plots) will be generated for each parameter and each cohort.

A summary table with the number and percentage of subjects with abnormally low, normal, and abnormally high values will be generated by measurement time, for each cohort.

Overall interpretation of echocardiograms will be listed by time point by cohort.

Graphs of actual mean(SE), mean of change from baseline(SE) by cohort over time will be plotted for mean ejection fraction.

Weight and BMI will be measured (see section  $\underline{12.1}$ ) for each cohort at the screening visit and at the completion visits.

Raw data and changes from baseline (Day 1) will be described by measurement time, for each cohort and listed.

Complete physical examination will be measured (see section 12.1) for each cohort at the screening visit, on Day 1, Week 1 and then once a week after.

Results from physical examination will be described by measurement time, for each cohort.

All physical examinations over time for any subject with any clinically significantly abnormal physical examinations will be listed as well as all individual data.

Pregnancy test will be performed (see section  $\underline{12.1}$ ) for each cohort at the screening visit and at the completion visits.

Positive pregnancy test will be listed as well as all individual data.

Toxicology testing will be listed.

# 9. Efficacy data

All efficacy analyses will be performed on the Safety set and, if necessary only, on the Per Protocol set.

# 9.1 Analysis Specifications

# 9.1.1 Level of Significance

No significance testing will be performed. However, a two-sided Clopper-Pearson 95% CI will be constructed around the proportion of subjects with SVRx and other virologic response parameters, for each cohort.

# 9.1.2 Data Handling Rules

Plasma HCV RNA values will be determined using the Roche Cobas Ampliprep/Cobas Taqman v2.0 assay with a lower limit of quantification (LLOQ) of 15 IU/mL and a limit of detection (LOD) of 15 IU/mL.

For the purpose of the analysis HCV RNA results "HCV RNA <15 IU/mL" will be imputed by LLOQ-1 IU/mL = 14 IU/mL before log transformation and "HCV RNA not detected" will be imputed by LOD-2 IU/mL= 13 IU/mL before log transformation.

# 9.2 Primary Efficacy Endpoint

The primary efficacy endpoint is sustained virologic response 12 weeks after the actual end of treatment (SVR12).

# 9.2.1 Definition

SVR12 is classified as success or failure according to the following algorithm based on HCV RNA values 12 weeks after the actual end of treatment.

**SVR12** is classified as a success (1) if at the time point of SVR12, HCV RNA value(s) meet one of the following:

- HCV RNA Not detected or
- < LLOQ detected and</li>
  - the sample is a confirmation\* visit or
  - the sample is the last available HCV RNA measurement or
  - at the next available measurement, HCV RNA not detected or HCV RNA < LLOQ detected
- $\geq$  LLOQ and
  - the sample is not from a confirmatory visit\* and
  - not the last available measurement in the study and
  - a next measurement is available and HCV RNA not detected or HCV RNA < LLOQ detected for this next measurement</li>

Otherwise SVR12 is classified as a failure (0).

\* Confirmed means that the criterion should be fulfilled at 2 or more consecutive time points or at the last observed time point.

# Time point of SVR12:

- o 12 weeks after the actual EOT (i.e. the last available measurement in the SVR12 analysis window)
- o or, if not available, the first available measurement at least 12 weeks after the actual EOT (i.e. the first available measurement after the SVR12 analysis window)
- o or, if not available (i.e. no measurement at least 12 weeks after the actual EOT), the subject is considered a failure.

# 9.2.2 Analysis Methods

The number and proportion of subjects with SVR12 will be tabulated overall and by cohort, a two-sided Clopper-Pearson 95% CI will be constructed.

# 9.3 Major Secondary Endpoints

Secondary efficacy endpoints include:

- Proportion of subjects with SVR4, SVR18 and SVR24
- Change from baseline in log<sub>10</sub> HCV RNA
- Actual values of log<sub>10</sub> HCV RNA
- Proportion of subjects with on-treatment virologic response at all timepoints (HCV RNA not detected; HCV RNA < LLOQ detected; HCV RNA not detected or HCV RNA < LLOQ detected)</li>
- Proportion of subjects with failure
- Proportion of subjects with on-treatment failure
- Proportion of subjects with viral relapse

#### 9.3.1 Definitions

**SVR4, SVR18 and SVR24** are defined similarly as SVR12 but with 4 weeks, 18 weeks and 24 weeks respectively, instead of 12 weeks.

In addition, for SVR24, the time point of SVR is defined as follows:

- o 24 weeks after actual EOT (i.e. the last available measurement in follow up Week 24 analysis window)
- o or, if not available, the first measurement available, after the follow-up Week 24 analysis window
- o or, if not available, the last measurement available in the SVR18 analysis window, on condition that the time point of SVR24 has been reached

- o or, if not available, the last measurement available in the follow up Week 12 analysis window (on condition that the time point of SVR24 has been reached)
- o or, if not available, the subject is considered as not having SVR24

For SVR18, the timepoint of SVR is defined as follows:

- o 18 weeks after the actual EOT (i.e. the last available measurement in follow up Week 18 analysis window)
- o or, if not available, the subject is considered as not having SVR18

**On-Treatment failure** is defined as subjects who did not achieve SVR12 and with confirmed HCV RNA  $\geq$ LLOQ at the actual end of study drug treatment. Includes subjects:

- With viral breakthrough, defined as a confirmed increase of >1 log10 in HCV RNA from nadir, or confirmed HCV RNA of >100 IU/mL in subjects whose HCV RNA had previously been <LLOQ while on treatment.
- With inadequate virologic response, defined as <1 log10 decline from baseline in HCV RNA after 4 weeks of treatment
- Who do not experience viral breakthrough or inadequate virologic response and have confirmed HCV RNA ≥LLOQ at the actual end of study drug treatment (e.g., completed study drug treatment, discontinued due to adverse events, withdrawal of consent).

# Viral Relapse is defined as follows:

Subjects who achieved HCV RNA <LLOQ at the actual end of study drug treatment and developed HCV RNA \geq LLOQ during post-treatment follow up.

Failure (No SVR12): Subjects who did not achieve SVR12, including:

- On-treatment failure (see above)
- Post-treatment failure, including subjects with:
  - Viral relapse (see above)
  - Missing HCV RNA at time point of SVR12

#### **On-treatment virologic response:**

Virologic response is quantitative HCV RNA concentration <LLOQ at any timepoint postfirst dose of study drug. An SVR is HCV RNA <LLOQ at Weeks 4, 8, 12, 18 or 24 after cessation of study treatment.

Time to virologic response is defined as the number of days since the first day of medication intake until the first day that the threshold was achieved. The following thresholds are considered:

- HCV RNA Not Detected
- HCV RNA Not Detected or HCV RNA < LLOQ Detected

### 9.3.2 Analysis Methods

The efficacy analysis will be performed on the Safety set and Per Protocol set, by cohort.

Descriptive statistics per cohort and per time point for the continuous parameter (actual values and changes from baseline in log<sub>10</sub> IU/mL HCV RNA) will be calculated.

Tabulations (numbers and proportions) per cohort and per time point for the categorical parameters will be provided. The observed proportion of subjects with SVR4 and SVR24 will be analyzed in the same way as the primary endpoint.

The influence of early virologic response parameters on SVR12 will be explored.

In addition, the reason for failure will be explored by type of failure (see definition of failure above). If more than one type of failure occurs, the order as presented below should be respected:

- a) viral relapse
- b) viral breakthrough
- c) confirmed detected at EOT
- d) missing at time point of SVR

Graphs of individual subject values (spaghetti plots) will be generated for each cohort for the viral load (VL) over time.

Graphs for mean VL change from baseline (+/- SD) over time will be generated for each cohort.

# 10. Reporting conventions

All tables, figures and listings are detailed in section 12.3. They will be prepared using SAS® software as rtf files and the rtf files will be compiled as Word files (one Word file by main section).

The footers will be presented as follows: --- STUDY <study protocol code> / <name of the program>.SAS / <name of the output>.RTF / DDMMMYY HH:MM ---.

Table and Listing Page Set Up Requirements:

- Font Type = Courier New
- Font Size = 8 pt (at a minimum)
- Page Margins: Top=2 cm; Bottom=2 cm; Left=2 cm; Right=2 cm
- Paper Size = A4 (21 cm x 29.7 cm)
- Page Orientation: Landscape
- Graphs: Portable Network Graphics (PNG) format

Summary statistics will be presented as follows.

| Parameter (unit) | Statistics<br>/ Category | Group X (N=xx) |
|------------------------|--------------------------|-------------------|
| Quantitative variable* | n | xx |
| | Mean ± SD | $xx.xx \pm xx.xx$ |
| | SEM | xx.xx |
| | Median | xx.xx |
| | Min ; Max | xx.x ; xx.x |
| Qualitative variable | Class 1 (n,%) | xx ( xx.x) |
| | Class 2 (n,%) | xx ( xx.x) |

<sup>\*</sup> For demographics and Baseline characteristics and for Safety summary tables:

All statistics, except the minimum and the maximum, will be provided with an additional decimal compared to the variable itself.

### For PK summary tables:

- if n=1 or n=2, do not display other statistics than n
- For tmax, only minimum, median, maximum and number of observations will be reported.
- For calculated values, PK parameters and descriptive statistics up to, but not including 100, display to 3 significant figures, for example:
  - 0.35769 is reported 0.358
  - 3.5769 is reported 3.58
  - 35.769 is reported 35.8
  - 357.69 is reported 358
  - For values  $\geq$  1000, the whole integer is reported (example 3576.9 is reported as 3577)

 $t_{max}$  and  $t_{lag}$  values are to be reported to 2 decimal places; half-life is to be reported to 1 decimal place.

Coefficient of Variation is reported to 1 decimal place.

Ratios and confidence interval are reported to 2 decimal places.

Drug concentration data that could not be obtained will be listed as NS (No Sample) in data tabulations.
# 11. Appendices

11.1 Appendix 1 - Schedule of assessments of the study

Table 6-1. Schedule of Events for 8 or 12\*-Week Treatment Groups

| Interval | | Day | | | | | | We | rek** | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Screen<br>-50 to -1 | 1 | 2 | 3 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| AL-335+ODV±SMV <sup>1</sup> | | < | | | | | | | | | | > |
| Obtain informed consent before study procedures | Х | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | |
| Height, Weight, BMI <sup>2</sup> | Х | | | | | | | | | | | X 2 |
| Drug Screen | Х | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | |
| Echocardiogram | X (=3 days) | | | | | | | X (+3 days) | | | | X (+3 days) |
| Triplicate 12-Lead electrocardiogram | X | Х | | | Х | Х | Х | X | X | Х | X | X |
| Physical Exam and vital signs 3 | Х | Х | | | Z | X | Х | Z | X | Х | X | Z |
| Hepatitis and HIV screen (HBsAg, HBsAB, HBcAb, HCVAb, HIVAb) | Х | | | | | | | | | | | |
| Alpha-fetoprotein, glycosylated HbA1C | X | | | | | | | | | | | |
| Liver Ultrasound (subjects with cirrhosis, if results from within the past 6 months are not available) | X | | | | | | | | | | | |
| HCV genotype | X | | | | | | | | | | | |
| IL28B genotype | | Х | | | | | | | | | | |
| Randomization <sup>4</sup> | | X | | | | | | | | | | |
| AE & Conmed Evaluation | Х | Х | Х | Х | Z | X | Х | X | Х | Х | Х | X |

Cohorts 1b, 2 to 16 may or may not include SMV. Dosing frequency will be qd except possibly for ODV which may also be dosed qod. Weight only collected at last treatment visit.

Complete Physical Exams, including vital signs (BP, HR, RR, body temperature), are to be done at screening, predose on Day 1, early termination, safety follow-up visits. Symptom directed physical exams and vitals are to be collected as necessary at all other visits.
 Randomization may take place up to 4 days before first dose.

Table 6-1. Schedule of Events for 8 or 12\*-Week Treatment Groups

| Interval | | Day | | | | | | W | eek** | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Screen<br>-50 to -1 | 1 | 2 | 3 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| PK Samples 5 | | Х | | | | Х | X | X | | Х | | X |
| Hematology <sup>6</sup> | X | Х | | | Х | Х | | X | | Х | | X |
| Serum Chemistries <sup>6</sup> | X | X | | | X | X | | X | | X | | X |
| Urinalysis | X | Х | | | Х | Х | | X | | X | | X |
| ALT/AST 6 | X | X | | | X | X | X | X | X | X | X | X |
| HCV RNA concentrations 7 | X | X | X | X | X | X | X | X | X | X | X | X |
| Plasma for drug resistance monitoring 8 | | Х | Х | Х | Х | X | X | X | X | X | X | X |
| Pregnancy Test 9 | X | | | | | | | X | | | | X |
| Stored serum sample 10 | X | Х | | | Х | Х | X | X | X | X | X | X |

<sup>&</sup>lt;sup>5</sup> A single predose PK sample will be collected at each indicated visit for AL-335 (and metabolites), ODV and SMV concentrations for all subjects. In addition, PK samples will be collected at Weeks 3 and 6, 2-4 hours postdose, and at Weeks 4 and 8, 6-8 hours postdose. Subjects in the intensive PK subset will have the following samples collected at the Week 2 visit Predose (within 0.5 hour) and 0.5, 1, 2, 3, 4, 6, 9, 12, and 24 hours postdose.

Blood for routine safety evaluations should be collected in a fasted state.

Plasma for HCV RNA analysis to be collected predose at Day 1.

Plasma collected for HCV RNA resistance monitoring will be collected at the same time as HCV RNA quantification. The Day 1 samples must be collected predose. Heterosexually active women of childbearing potential. A highly sensitive pregnancy test (e.g., urine or plasma) must be conducted immediately (within 4 days) prior to initiating treatment on Day 1 (local results may be used for this eligibility determination)

For additional safety investigations as needed.

<sup>\*</sup>If a 12-week regimen is evaluated, the Week 5, 6, 7, and 8 visits will be repeated at Weeks 9, 10, 11, and 12, respectively.

<sup>\*\*</sup> Weekly visit may occur ±1 day from the expected visit date.

Table 6-2. Schedule of Events for a 6-Week Treatment Group

| Interval | | Day | | | | | | Week* | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Screen<br>-50 to -1 | 1 | 2 | 3 | 1 | 2 | 3 | 4 | 5 | 6 |
| AL-335+ODV±SMV <sup>1</sup> | | < | | | | | | | | ·> |
| Obtain informed consent before study procedures | X | | | | | | | | | |
| Demographics | Х | | | | | | | | | |
| Height, Weight, BMI <sup>2</sup> | X | | | | | | | | | X² |
| Drug Screen | X | | | | | | | | | |
| Medical History | X | | | | | | | | | |
| Echocardiogram | X (±3 days) | | | | | | | X (±3 days) | | X (±3 days) |
| Triplicate 12-Lead electrocardiogram | X | X | | | X | X | Х | X | X | X |
| Physical Exam and vital signs <sup>3</sup> | X | X | | | X | Х | Х | X | X | X |
| Hepatitis and HIV screen (HBsAg, HBsAB, HBcAb, HCVAb, HIVAb) | X | | | | | | | | | |
| Alpha-fetoprotein, glycosylated HbA1C | X | | | | | | | | | |
| Liver Ultrasound (subjects with cirrhosis, if results from within the past 6 months are not available) | X | | | | | | | | | |
| HCV genotype | X | | | | | | | | | |
| IL28B genotype | | X | | | | | | | | |
| Randomization <sup>4</sup> | | X | | | | | | | | |
| AE & Conmed Evaluation | X | Х | Х | X | Х | Х | Х | X | Х | Х |

<sup>&</sup>lt;sup>1</sup> Cohorts 1b, 2 to 16 may or may not include SMV. Dosing frequency will be qd except possibly for ODV which may also be dosed qod.

Weight only collected at Week 6.
 Complete Physical Exams, including vital signs (BP, HR, RR, body temperature), are to be done at screening, predose on Day 1, early termination, safety follow-up visits. Symptom directed physical exams and vitals are to be collected as necessary at all other visits.
 Randomization may take place up to 4 days before first dose.

Table 6-2. Schedule of Events for a 6-Week Treatment Group

| Interval | | Day | | | | | | Week* | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Screen<br>-50 to -1 | 1 | 2 | 3 | 1 | 2 | 3 | 4 | 5 | 6 |
| PK Samples <sup>5</sup> | | X | | | | Х | Х | X | | X |
| Hematology <sup>6</sup> | X | X | | | X | X | | X | | X |
| Serum Chemistries <sup>6</sup> | X | X | | | X | Х | | X | | X |
| Urinalysis | X | X | | | X | X | | X | | X |
| ALT/AST 6 | X | X | | | X | Х | X | X | X | X |
| HCV RNA concentrations 7 | X | X | X | X | X | Х | Х | X | X | X |
| Plasma for drug resistance monitoring 8 | | X | X | X | X | X | X | X | X | X |
| Pregnancy Test 9 | X | | | | | | | X | | |
| Stored serum sample 10 | X | X | | | Х | Х | Х | X | Х | X |

<sup>&</sup>lt;sup>5</sup> A single predose PK sample will be collected at each indicated visit for AL-335(and metabolites), ODV and SMV concentrations for all subjects. In addition, PK samples will be collected at Weeks 3 and 6, 2-4 hours postdose, and at Week 4, 6-8 hours postdose. Subjects in the intensive PK subset will have the following samples collected at the Week 2 visit Predose (within 0.5 hour) and 0.5, 1, 2, 3, 4, 6, 9, 12, and 24 hours postdose.

Blood for routine safety evaluations should be collected in a fasted state.

Plasma for HCV RNA analysis to be collected predose at Day 1.

Plasma collected for HCV RNA resistance monitoring will be collected at the same time as HCV RNA quantification. The Day 1 samples must be collected predose.

<sup>9</sup> A highly sensitive pregnancy test (e.g., urine or plasma) must be conducted immediately (within 4 days) prior to initiating treatment on Day 1 (local results may be used for this eligibility determination)

10 For additional safety investigations as needed.

\* Weekly visit may occur ±1 day from the expected visit date.

Table 6-3. Schedule of Events for a 4-Week Treatment Group

| Interval | Screen | Day 1 | Day 2 | Day 3 | Week 1* | Week 2* | Week 3* | Week 4* |
|---|---|---|---|---|---|---|---|---|
| Assessments | -50 to -1 | · | • | • | | | | |
| AL-335+ODV±SMV <sup>1</sup> | | << | | | | | | > |
| Obtain informed consent before study procedures | X | | | | | | | |
| Demographics | X | | | | | | | |
| Height, Weight, BMI <sup>2</sup> | Х | | | | | | | X 2 |
| Drug Screen | X | | | | | | | |
| Medical History | X | | | | | | | |
| Echocardiogram | X (+3 days) | | | | | | | X (+3 days) |
| Triplicate 12-Lead electrocardiogram | X | X | | | X | X | Z | X |
| Physical Exam and vital signs 3 | X | X | | | X | X | X | X |
| Hepatitis and HIV screen (HBsAg, HBsAB,<br>HBcAb, HCVAb, HIVAb) | X | | | | | | | |
| Alpha-fetoprotein, glycosylated HbA1C | X | | | | | | | |
| Liver Ultrasound (subjects with cirrhosis, if results from within the past 6 months are not available) | Х | | | | | | | |
| HCV genotype/subtype | X | | | | | | | |
| IL28B genotype | | X | | | | | | |
| Randomization <sup>4</sup> | | X | | | | | | |
| AE & Conmed Evaluation | X | X | X | X | X | Х | Х | X |

<sup>&</sup>lt;sup>1</sup> Cohorts 1b, 2 to 16 may or may not include SMV. Dosing frequency will be qd except possibly for ODV which may also be dosed qod.

Weight only collected at Week 4.
 Complete Physical Exams, including vital signs (BP, HR, RR, body temperature), are to be done at screening, predose on Day 1, early termination, safety follow-up visits. Symptom directed physical exams and vitals are to be collected as necessary at all other visits. Vital signs will be collected at all visits indicated.
 Randomization may take place up to 4 days before first dose.

Table 6-3. Schedule of Events for a 4-Week Treatment Group

| Assessments | Screen<br>-50 to -1 | Day 1 | Day 2 | Day 3 | Week 1* | Week 2* | Week 3* | Week 4* |
|---|---|---|---|---|---|---|---|---|
| PK Samples 5 | | X | | | X | X | X | X |
| Hematology <sup>6</sup> | X | X | | | X | X | | X |
| Serum Chemistries <sup>6</sup> | X | X | | | X | X | | X |
| Urinalysis | X | X | | | X | X | | X |
| ALT/AST 6 | X | X | | | X | Х | X | X |
| HCV RNA concentrations 7 | X | X | Х | X | X | X | X | X |
| Plasma for drug resistance monitoring 8 | | X | Х | X | Х | X | X | X |
| Pregnancy Test 9 | X | | | | | | | X |
| Stored serum sample 10 | X | X | | | X | X | X | X |

A single predose PK sample will be collected at each indicated visit for AL-335 (and metabolites), ODV and SMV concentrations for all subjects. In addition, PK samples will be collected at Week 3, 2-4 hours postdose, and at Week 4, 6-8 hours postdose. Subjects in the intensive PK subset will have the following samples collected at the Week 2 visit Predose (within 0.5 hour) and 0.5, 1, 2, 3, 4, 6, 9, 12, and 24 hours postdose.

Blood for routine safety evaluations should be collected in a fasted state.

Plasma for HCV RNA analysis to be collected predose at Day 1, 2 and 3.
Plasma collected for HCV RNA resistance monitoring will be collected at the same time as HCV RNA quantification. The Day 1 samples must be collected predose.

A highly sensitive pregnancy test (e.g., urine or plasma) must be conducted immediately (within 4 days) prior to initiating treatment on Day 1 (local results may be used for this eligibility determination)
 For additional safety investigations as needed.
 \* Weekly visit may occur ±1 day from the expected visit date.

Table 6-4. Schedule of Events for Post-dosing (Safety and Virology) Follow-up Visits (All Treatment Cohorts)

| Post-dosing Follow-up | Post-dosing Follow-up | | | | | | |
|---|---|---|---|---|---|---|---|
| | Early | Safety Follow-up Visit<br>4 Weeks (±1 week) | Virology Fo | reatment <sup>2</sup> OR<br>earlier]) <sup>3</sup> | | | |
| Assessment | Termination<br>(ET) Visit <sup>1</sup> | After the Last Actual<br>Dose of Study Drug | Week 4<br>(±1 week) <sup>4</sup> | Week 8<br>(±1 weeks) | Week 12<br>(±2 weeks) | Week 18<br>(±2 weeks) | Week 24<br>(±2 weeks) |
| Physical Exam <sup>5</sup> | X | X | | | | | |
| Echocardiogram | X | X | | | | | |
| Vital Signs | X | X | | | | | |
| Triplicate 12 Lead ECG | X | X | | | | | |
| Serum Chemistry w/ ALT & AST | X | X | | | | | |
| Hematology | X | X | | | | | |
| Urinalysis | X | X | | | | | |
| HCV RNA concentration | X | X | X | X | X | X | X |
| Plasma for drug resistance monitoring | X | X | X | X | X | X | X |
| AE & Conmed Evaluation | X | X | X | X | X | X | X |
| PK Samples 6 | X | X | X | X | X | X | X |
| Pregnancy test <sup>7</sup> | X | X | | X | X | | X |
| Stored Serum Sample <sup>8</sup> | X | X | | | | | |

Subjects who prematurely discontinue from their assigned study treatment should return to the clinic as soon as possible for an Early Termination Visit. If the timing of the Early Termination Visit coincides with the Safety Follow up Visit, then assessments for the Early Termination Visit should be conducted.

<sup>2</sup> For subjects with less than lower limit of quantitation (<LLOQ) HCV RNA at actual end of treatment (EOT) (if prematurely discontinued treatment, discontinuation was for reasons other than on-treatment virologic failure (e.g., AE).

On-treatment failure is defined as virologic failure or breakthrough. No subject will be followed for more than 24 weeks.

<sup>4</sup> Note: The Week 4 Virology Follow up Visit will coincide with the Safety Follow-up Visit for most subjects and may be replaced by the Safety Follow-up Visit in these cases; it will not coincide for subjects who have relapse or for subjects who discontinue early with <LLOQ HCV RNA.

<sup>5</sup> Complete Physical Exams, including vital signs (BP, HR, RR, body temperature), are to be done at screening, predose on Day 1, early termination, safety follow-up visits. Symptom directed physical exams and vitals are to be collected as necessary at all other visits.

PK sampling will be conducted for ODV at the time of visit.

Heterosexually active women of childbearing potential.

For additional safety investigations as needed.

## 11.2 Appendix 2 - Criteria for Potentially Clinically Significant Abnormalities (PCSA)

| Vital signs | | |
|---|---|---|
| PR | ≤ 50 bpm | ≥ 120 bpm |
| SBP | ≤ 90 mmHg | > 140 mmHg |
| DBP | ≤ 50 mmHg | > 90 mmHg |
| ECG parameters | | |
| PR | <120 ms | > 200 ms |
| QRS | | > 120 ms |
| QTcB or QTcF | | $> 450 - \le 480 \text{ ms}$ |
| | | > 480 ms |
| | | > 500 ms |
| | | change from baseline $\geq 30 - \leq 60 \text{ ms}$ |
| | | change from baseline > 60 ms |

11.3 Appendix 3 - List of tables, listings and figures included in the clinical study report

| NUMBER | TITLE |
|---|---|
| 14 | Tables, figures and graphs referred to but not included in the text |
| 14.1 | Demographic data |
| 14.1.1 | Description of study subjects |
| 14.1.1.1 | Subjects disposition - Included set |
| 14.1.1.2 | Analysis sets – Included set |
| 14.1.2 | Protocol deviations |
| 14.1.2.1 | Deviations relating to inclusion/exclusion criteria - Safety set |
| 14.1.2.2 | Other deviations - Safety set |
| 14.1.3 | Demographic data and baseline characteristics |
| 14.1.3.1.1 | Demographic data - Safety set |
| 14.1.3.1.2 | Demographic data - PKS |
| 14.1.3.2 | Other baseline characteristics |
| 14.1.3.2.1.1 | HCV genotype – Safety set |
| 14.1.3.2.1.2 | HCV genotype – PKS |
| 14.1.3.2.2.1 | HCV RNA – Safety set |
| 14.1.3.2.2.2 | HCV RNA – PKS |
| 14.1.3.2.3.1 | Serology - Safety set |
| 14.1.3.2.3.2 | Serology - PKS |
| 14.1.3.2.4 | Listing of positive results of serology - Safety set |
| 14.1.3.2.5.1 | Cirrhosis status - Safety set |
| 14.1.3.2.5.2 | Cirrhosis status - PKS set |
| 14.1.3.2.6.1 | Liver biopsy – Safety set |

| 14.1.3.2.6.2 | Liver biopsy – PKS |
|---|---|
| 14.1.3.2.7.1 | Fibroscan - Safety set |
| 14.1.3.2.7.2 | Fibroscan - PKS set |
| 14.1.3.3 | Medical and surgical history |
| 14.1.3.3.1 | Previous medical and surgical history (except liver diseases) - Safety set |
| 14.1.3.3.2 | Ongoing medical and surgical history (except liver diseases) - Safety set |
| 14.1.3.3.3 | Previous liver diseases - Safety set |
| 14.1.3.3.4 | Ongoing liver diseases - Safety set |
| 14.1.3.4 | Previous and concomitant medications |
| 14.1.3.4.1 | Previous medications - Safety set |
| 14.1.3.4.2 | Concomitant medications - Safety set |
| 14.2 | Pharmacokinetic data |
| 14.2.1 | Plasma concentrations |
| 14.2.1.1 | AL-335, ALS-022399 and ALS-022227 |
| 14.2.1.1.1 | Plasma concentrations for AL-335, ALS-022399 and ALS-022227 -<br>Pharmacokinetic set |
| 14.2.1.1.2 | Graphs of plasma concentrations means (±SD) over time for AL-335, ALS-022399 and ALS-022227 - Pharmacokinetic set |
| 14.2.1.1.2.1 | Graphs of plasma concentrations means (±SD) over time for AL-335, ALS-022399 and ALS-022227 by analyte |
| 14.2.1.1.2.2 | Graphs of plasma concentrations means (±SD) over time for AL-335, ALS-022399 and ALS-022227 by cohort |
| 14.2.1.1.3 | Graphs of trough plasma concentrations means (±SD) over time for AL-335, ALS-022399 and ALS-022227 - Pharmacokinetic set |

| 14.2.1.2 | Simeprevir |
|---|---|
| 14.2.1.2.1 | Plasma concentrations for simeprevir - Pharmacokinetic set |
| 14.2.1.2.2 | Graphs of plasma concentrations means (±SD) over time for simeprevir - Pharmacokinetic set |
| 14.2.1.2.3 | Graphs of trough plasma concentrations means (±SD) over time for simeprevir - Pharmacokinetic set |
| 14.2.1.3 | Odalasvir |
| 14.2.1.3.1 | Plasma concentrations for odalasvir - Pharmacokinetic set |
| 14.2.1.3.2 | Graphs of plasma concentrations means (±SD) over time for odalasvir - Pharmacokinetic set |
| 14.2.1.3.3 | Graphs of trough plasma concentrations means (±SD) over time for odalasvir - Pharmacokinetic set |
| 14.2.2 | PK parameters in plasma |
| 14.2.2.1 | AL-335, ALS-022399 and ALS-022227 |
| 14.2.2.1.1 | PK parameters in plasma for AL-335, ALS-022399 and ALS-022227 - Pharmacokinetic set |
| 14.2.2.1.2 | Scatter plots of $C_{max}$ and $AUC_{0-\tau}$ for AL-335, ALS-022399 and ALS-022227 by cohort - Pharmacokinetic set |
| 14.2.2.1.3 | Box whisker plots of $C_{max}$ and $AUC_{0-\tau}$ for AL-335, ALS-022399 and ALS-022227 by cohort - Pharmacokinetic set |
| 14.2.2.2 | Simeprevir |
| 14.2.2.2.1 | PK parameters in plasma for simeprevir - Pharmacokinetic set |
| 14.2.2.2.2 | Scatter plots of $C_{\text{max}}$ and $AUC_{0\text{-}\tau}$ for simeprevir by cohort - Pharmacokinetic set |
| 14.2.2.2.3 | Box whisker plots of $C_{\text{max}}$ and $AUC_{0-\tau}$ for simeprevir by cohort - Pharmacokinetic set |
| 14.2.2.3 | Odalasvir |

| 14.2.2.3.1 | PK parameters in plasma for odalasvir - Pharmacokinetic set |
|---|---|
| 14.2.2.3.2 | Scatter plots of $C_{\text{max}}$ and $AUC_{0-\tau}$ for odalasvir by cohort - Pharmacokinetic set |
| 14.2.2.3.3 | Box whisker plots of $C_{\text{max}}$ and $AUC_{0-\tau}$ for odalasvir by cohort - Pharmacokinetic set |
| 14.3 | Safety data |
| 14.3.1 | Adverse events |
| 14.3.1.1 | Adverse events - Safety set |
| 14.3.1.2 | Treatment emergent adverse events |
| 14.3.1.2.1 | Treatment emergent adverse events summary table - Safety set |
| 14.3.1.2.2 | Treatment emergent adverse events - Safety set |
| 14.3.1.2.3 | Treatment emergent adverse events by preferred term - Safety set |
| 14.3.1.2.4 | Treatment emergent adverse events by intensity - Safety set |
| 14.3.1.2.5 | Treatment emergent adverse events by causality - Safety set |
| 14.3.1.2.6 | Treatment emergent serious adverse events by preferred term - Safety set |
| 14.3.1.2.7 | Treatment emergent adverse events leading to any study drug discontinuation by preferred term - Safety set |
| 14.3.1.2.8 | Treatment emergent adverse events of special interest - Safety set |
| 14.3.1.2.9 | Adverse Events with fatal outcome – Included set |
| 14.3.1.2.10 | The incidence and comparable prevalence rate per 2-week time interval for any AEs |
| 14.3.1.2.11 | The incidence rates for adverse events of special interest by WHO toxicity grade |
| 14.3.1.2.12 | The incidence rates for adverse events of special interest by relationship to study drugs |

| 14.3.1.2.13 | The incidence rates for serious adverse events of special interest by relationship to study drugs |
|---|---|
| 14.3.1.2.14 | Time to the first occurrence of adverse events of special interest |
| 14.3.1.2.15 | The incidence and comparable prevalence rate per 2-week time interval for adverse events of special interest |
| 14.3.1.3.1 | Graph of incidence and comparable prevalence rate for any AE over time |
| 14.3.1.3.2 | Kaplan Meier Curve for the Time to Onset of adverse events of special interest |
| 14.3.1.3.3 | Graph of incidence and comparable prevalence rate for adverse event of special interest over time |
| 14.3.1.3.4 | Bar chart of the worst toxicity grade of cardiac events over time |
| 14.3.2.1 | Listing of deaths, SAEs and TEAEs leading to study drug discontinuation - Safety set |
| 14.3.2.2 | Listing of TEAEs with grade 3 or grade 4 - Safety set |
| 14.3.2.3 | Glossary of adverse events |
| 14.3.2.4 | Listing of adverse events for subjects who met the study stopping rules |
| 14.3.3 | Clinical laboratory data |
| 14.3.3.1 | Haematology |
| 14.3.3.1.1 | Haematology parameters - Safety set |
| 14.3.3.1.2 | Number and percentage of subjects by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) – Worst post-baseline value - Safety set |
| 14.3.3.1.3 | Number and percentage of subjects by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) – By measurement time - Safety set |
| 14.3.3.1.4 | Listing of all values for subjects presenting any treatment emergent value that is grade 3 and 4 (toxicity grading scale) - Safety set |
| 14.3.3.1.5 | Listing of subjects with treatment emergent abnormal values - |

| | Safety set |
|---|---|
| 14.3.3.1.6 | Graphs of individual subject values (spaghetti plots) – Safety Set |
| 14.3.3.1.7 | Cross-tabulation of the worst toxicity grades versus baseline |
| 14.3.3.1.8 | Plot of mean(SE) by cohort over time |
| 14.3.3.1.9 | Plot of mean(SE) change from baseline by cohort over time |
| 14.3.3.1.10 | Bar chart of the treatment emergent abnormality by toxicity grade over time |
| 14.3.3.2 | Blood chemistry |
| 14.3.3.2.1 | Blood chemistry parameters - Safety set |
| 14.3.3.2.2 | Number and percentage of subjects by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) – Worst post-baseline value - Safety set |
| 14.3.3.2.3 | Number and percentage of subjects by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) – By measurement time - Safety set |
| 14.3.3.2.4 | Listing of all values for subjects presenting any treatment emergent values that are grade 3 and 4 (toxicity grading scale) - Safety set |
| 14.3.3.2.5 | Listing of subjects with treatment emergent abnormal values -<br>Safety set |
| 14.3.3.2.6 | Graphs of individual subject values (spaghetti plots) – Safety Set |
| 14.3.3.2.7 | Cross-tabulation of the worst toxicity grades versus baseline |
| 14.3.3.2.8 | Plot of mean(SE) by cohort over time |
| 14.3.3.2.9 | Plot of mean(SE) change from baseline by cohort over time |
| 14.3.3.2.10 | Bar chart of the treatment emergent abnormality by toxicity grade over time |
| 14.3.3.3 | Coagulation - Safety set |
| 14.3.3.3.1 | Coagulation parameters - Safety set |
| 14.3.3.3.2 | Number and percentage of subjects by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) – Worst post-baseline value - Safety set |

| 14.3.3.3.3 | Number and percentage of subjects by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) – By measurement time - Safety set |
|---|---|
| 14.3.3.3.4 | Listing of all values for subjects presenting any treatment emergent values that are grade 3 and 4 (toxicity grading scale) - Safety set |
| 14.3.3.3.5 | Listing of subjects with treatment emergent abnormal values -<br>Safety set |
| 14.3.3.3.6 | Cross-tabulation of the worst toxicity grades versus baseline |
| 14.3.3.3.7 | Plot of mean(SE) by cohort over time |
| 14.3.3.3.8 | Plot of mean(SE) change from baseline by cohort over time |
| 14.3.3.3.9 | Bar chart of the treatment emergent abnormality by toxicity grade over time |
| 14.3.3.4 | Urinalysis - Safety set |
| 14.3.3.4.1 | Urinalysis parameters - Safety set |
| 14.3.3.4.2 | Number and percentage of subjects by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) – Worst post-baseline value - Safety set |
| 14.3.3.4.3 | Number and percentage of subjects by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) – By measurement time - Safety set |
| 14.3.3.4.4 | Listing of all values for subjects presenting any treatment emergent values that are grade 3 and 4 (toxicity grading scale) - Safety set |
| 14.3.3.4.5 | Listing of subjects with treatment emergent abnormal values -<br>Safety set |
| 14.3.4 | Other safety parameters |
| 14.3.4.1 | Vital signs data |
| 14.3.4.1.1 | Vital signs parameters - Safety set |
| 14.3.4.1.2 | Number and percentage of subjects presenting PCSA values - Safety set |
| 14.3.4.1.3 | Listing of subjects presenting PCSA values - Safety set |

| 14.3.4.1.4 | Number and percentage of subjects presenting abnormal values – Worst post-baseline value - Safety set |
|---|---|
| 14.3.4.1.5 | Number and percentage of subjects presenting abnormal values – By measurement time - Safety set |
| 14.3.4.1.6 | Listing of subjects presenting abnormal values - Safety set |
| 14.3.4.1.7 | Plots of mean (SE) by cohort over time |
| 14.3.4.2 | Electrocardiogram data |
| 14.3.4.2.1 | ECG parameters – Safety set |
| 14.3.4.2.2 | Number and percentage of subjects with PCSA values - Safety set |
| 14.3.4.2.3 | Listing of subjects presenting PCSA values - Safety set |
| 14.3.4.2.4 | Listing of All ECG Parameters over time for Subjects with Any Post-<br>baseline Overall Statement of Potentially Clinically Significant<br>Abnormal ECG |
| 14.3.4.2.5 | Listing of Subjects with Potentially Progressive PR Prolongation |
| 14.3.4.2.6 | Number and percentage of subjects presenting abnormal values – Worst post-baseline value - Safety set |
| 14.3.4.2.7 | Number and percentage of subjects presenting abnormal values – By measurement time - Safety set |
| 14.3.4.2.8 | Listing of subjects presenting abnormal values - Safety set |
| 14.3.4.2.9 | Graphs of individual subject values (spaghetti plots) – Safety Set |
| 14.3.4.2.10 | Cross-Tabulation of the worst ECG abnormalities in actual value versus the baseline value |
| 14.3.4.2.11 | Cross-Tabulation of the worst QTc increase versus the abnormality on the actual value |
| 14.3.4.2.12 | Plots of actual mean(SE) by cohort over time |
| 14.3.4.2.13 | Plots of mean change from baseline(SE) by cohort over time |
| 14.3.4.2.14 | Spaghetti plot of PR for the patients who had prolonged PR interval |

| | or AV block (grade>=1) |
|---|---|
| 14.3.4.3 | Echocardiogram data |
| 14.3.4.3.1 | Summary Table of Maximum Decrease from baseline in Mean<br>Ejection Fraction – Safety set |
| 14.3.4.3.2 | Number and Percentage of subjects who have a decrease greater han 5% or ≤10% and >10% compared to baseline – Safety set |
| 14.3.4.3.3 | Listing of all EF values for Subjects with any >5%-≤10 Decrease from baseline in Mean Ejection Fraction – Safety set |
| 14.3.4.3.4 | Listing of all EF values for Subjects with any More Than 10%<br>Decrease from baseline in Mean Ejection Fraction – Safety set |
| 14.3.4.3.5 | Listing of Ejection Fraction Data and Overall Comment – Safety set |
| 14.3.4.3.6 | Echocardiogram parameters – Safety set |
| 14.3.4.3.7 | Number and percentage of subjects with abnormal values - Safety set |
| 14.3.4.3.8 | Graphs of individual subject values (spaghetti plots) – Safety set |
| 14.3.4.3.9 | Plots of actual mean(SE) by cohort over time |
| 14.3.4.3.10 | Plots of mean change from baseline(SE) by cohort over time |
| 14.3.4.4 | Weight and BMI – Safety set |
| 14.3.4.5 | Physical examination |
| 14.3.4.5.1 | Physical examination - Safety set |
| 14.3.4.5.2 | Abnormal physical examination - Safety set |
| 14.3.4.6 | Positive pregnancy test - Safety set |
| 14.4 | Efficacy data |
| 14.4.1 | HCV RNA – Safety set |
| 14.4.2 | Number and percentage of subjects who are HCV RNA not detected or below the limit of quantification – Safety set |

| 14.4.3 | Sustained virologic response |
|---|---|
| 14.4.3.1 | Number and percentage of subjects with sustained virologic response 12 weeks after end of treatment – Safety set |
| 14.4.3.2 | Number and percentage of subjects with sustained virologic response 4 weeks after end of treatment – Safety set |
| 14.4.3.3 | Number and percentage of subjects with sustained virologic response 24 weeks after end of treatment – Safety set |
| 14.4.4 | Number and percentage of subjects with virologic failure – Safety set |
| 14.4.5.1 | Graphs of individual subject values of viral load (spaghetti plots) – Safety set |
| 14.4.5.2 | Graphs of mean viral load change from baseline – Safety set |
| 16.2 | SUBJECT DATA LISTINGS |
| 16.2.1 | Subjects disposition |
| 16.2.1.1 | Discontinued subjects - Included set |
| 16.2.1.2 | Subjects disposition and analysis sets - Included set |
| 16.2.1.3 | End of study status - Included set |
| 16.2.1.4 | Subject visit dates - Included set |
| 16.2.2 | Protocol deviations |
| 16.2.2.1 | Deviations relating to inclusion/exclusion criteria - Safety set |
| 16.2.2.2 | Other deviations – Safety set |
| 16.2.3 | Subjects excluded from analysis sets - Included set |
| 16.2.4 | Demographic data and baseline characteristics |
| 16.2.4.1 | Demographic data and baseline characteristics - Safety set |
| 16.2.4.2 | Other baseline characteristics |
| 16.2.4.2.1 | HCV genotype – Safety set |

| 16.2.4.2.2 | HCV RNA – Safety set |
|---|---|
| | · |
| 16.2.4.2.3 | Serology - Safety set |
| 16.2.4.2.4 | Childbearing status – Safety set |
| 16.2.4.2.5 | Contraception method – Safety set |
| 16.2.4.2.6 | Alcohol consumption – Safety set |
| 16.2.4.2.7 | Cirrhosis status – Safety set |
| 16.2.4.2.8 | Liver biopsy – Safety set |
| 16.2.4.2.9 | Fibroscan – Safety set |
| 16.2.4.2.10 | Child-Pugh class assessment (only for compensated cirrhosis cohort) – Safety set |
| 16.2.4.2.11 | patocellular carcinoma assessment (only for compensated<br>rhosis cohorts) – Safety set |
| 16.2.4.3 | Medical and surgical history |
| 16.2.4.3.1 | Medical and surgical history (except liver diseases) – Safety set |
| 16.2.4.3.2 | Liver diseases – Safety set |
| 16.2.4.4 | Previous and concomitant medications |
| 16.2.4.4.1 | Previous medications - Safety set |
| 16.2.4.4.2 | Concomitant medications - Safety set |
| 16.2.5 | Compliance and/or drug concentration data |
| 16.2.5.1 | Compliance and dosing data |
| 16.2.5.1.1 | IMP administration – Safety set |
| 16.2.5.1.2 | Meals intake – Safety set |
| 16.2.5.2 | Pharmacokinetic data |
| 16.2.5.2.1 | Plasma pharmacokinetic concentrations and parameters |
| 16.2.5.2.1.1 | AL-335, ALS-022399 and ALS-022227 |

| 16.2.5.2.1.1.1 | Plasma concentrations for AL-335, ALS-022399 and ALS-022227 -<br>Pharmacokinetic set |
|---|---|
| 16.2.5.2.1.1.2 | Plasma concentrations for AL-335, ALS-022399 and ALS-022227 — Subgroup of subjects who discontinue the study for an adverse event, experience a severe adverse event or a serious adverse event - Pharmacokinetic set |
| 16.2.5.2.1.1.3 | Individual plasma concentration time curves for AL-335, ALS-022399 and ALS-022227- Pharmacokinetic set |
| 16.2.5.2.1.1.4 | PK parameters in plasma for AL-335, ALS-022399 and ALS-022227 - Pharmacokinetic set |
| 16.2.5.2.1.1.5 | PK parameters in plasma for AL-335, ALS-022399 and ALS-022227 – Subgroup of subjects who discontinue the study for an adverse event, experience a severe adverse event or a serious adverse event – Pharmacokinetic set |
| 16.2.5.2.1.2 | Simeprevir |
| 16.2.5.2.1.2.1 | Plasma concentrations for Simeprevir - Pharmacokinetic set |
| 16.2.5.2.1.2.2 | Plasma concentrations for Simeprevir – Subgroup of subjects who discontinue the study for an adverse event, experience a severe adverse event or a serious adverse event - Pharmacokinetic set |
| 16.2.5.2.1.2.3 | Individual plasma concentration time curves for Simeprevir -<br>Pharmacokinetic set |
| 16.2.5.2.1.2.4 | PK parameters in plasma for Simeprevir - Pharmacokinetic set |
| 16.2.5.2.1.2.5 | PK parameters in plasma for Simeprevir – Subgroup of subjects who discontinue the study for an adverse event, experience a severe adverse event or a serious adverse event - Pharmacokinetic set |
| 16.2.5.2.1.3 | Odalasvir |
| 16.2.5.2.1.3.1 | Plasma concentrations for Odalasvir - Pharmacokinetic set |
| 16.2.5.2.1.3.2 | Plasma concentrations for Odalasvir – Subgroup of subjects who discontinue the study for an adverse event, experience a severe adverse event or a serious adverse event - Pharmacokinetic set |

| 16.2.5.2.1.3.3 | Individual plasma concentration time curves for Odalasvir -<br>Pharmacokinetic set |
|---|---|
| 16.2.5.2.1.3.4 | PK parameters in plasma for Odalasvir - Pharmacokinetic set |
| 16.2.5.2.1.3.5 | PK parameters in plasma for Odalasvir – Subgroup of subjects who discontinue the study for an adverse event, experience a severe adverse event or a serious adverse event - Pharmacokinetic set |
| 16.2.6 | Efficacy data |
| 16.2.6.1 | HCV RNA – Safety set |
| 16.2.6.2 | HCV RNA for subjects with virologic failures— Safety set |
| 16.2.7 | Adverse event listings |
| 16.2.7.1 | All adverse events – Included set |
| 16.2.7.2 | Treatment emergent adverse events - Safety set |
| 16.2.7.3 | Serious adverse events – Included set |
| 16.2.7.4 | Treatment emergent adverse events leading to study drug discontinuation – Safety set |
| 16.2.7.5 | Treatment emergent adverse events of special interest - Safety set |
| 16.2.7.6 | Adverse events with fatal outcome – Included set |
| 16.2.7.7 | Rash assessments |
| 16.2.7.7.1 | Photosensitivity – Safety set |
| 16.2.7.7.2 | Rash assessments – Safety set |
| 16.2.7.7.3 | Associated rash or cutaneous event – Safety set |
| 16.2.7.7.4 | Rash or cutaneous event follow-up – Safety set |
| 16.2.7.7.5 | Final rash, cutaneous event or photosensitivity evaluation – Safety set |
| 16.2.7.7.6 | Primary lesions of rash or cutaneous event – Safety set |
| 16.2.7.7.7 | Secondary lesions of rash or cutaneous event – Safety set |

| 16.2.7.7.8 | Rash questionnaire – Safety set |
|---|---|
| 16.2.7.7.9 | Rash event grading – Safety set |
| 16.2.8 | Clinical laboratory data |
| 16.2.8.1 | Haematology |
| 16.2.8.1.1 | Normal ranges for SI units and local units |
| 16.2.8.1.2 | All haematology values (SI unit) - Safety set |
| 16.2.8.2 | Blood chemistry |
| 16.2.8.2.1 | Normal ranges for SI units and local units |
| 16.2.8.2.2 | All blood chemistry values (SI unit) - Safety set |
| 16.2.8.3 | Coagulation |
| 16.2.8.3.1 | Normal ranges for SI units and local units |
| 16.2.8.3.2 | All coagulation values (SI unit) - Safety set |
| 16.2.8.4 | Urinalysis |
| 16.2.8.4.1 | Normal ranges for SI units and local units |
| 16.2.8.4.2 | All urinalysis values (SI unit) - Safety set |
| 16.2.8.5 | Hormonology – Safety set |
| 16.2.9 | Other safety parameters |
| 16.2.9.1 | Vital signs data |
| 16.2.9.1.1 | PCSA ranges |
| 16.2.9.1.2 | Vital signs parameters - Safety set |
| 16.2.9.2 | Electrocardiogram data |
| 16.2.9.2.1 | PCSA ranges |
| 16.2.9.2.2.1 | Standard 12-lead ECG parameters (centrally read data) - Safety set |

| 16.2.9.3 | Echocardiogram data – Safety set |
|----------|-----------------------------------|
| 16.2.9.4 | Weight and BMI – Safety set |
| 16.2.9.5 | Physical examination – Safety set |
| 16.2.9.6 | Pregnancy test - Safety set |
| 16.2.9.7 | Toxicology – Safety set |

### 11.4 Appendix 4: Events of special/clinical interest

# 11.4.1 Search terms for Events of Special/Clinical Interest

| | MedrDRA | Searching Terms |
|---|---|---|
| | Term Level | |
| Events of special interest | | |
| - | G) (0 | |
| Cardiac Events | SMQ | Cardiac arrhythmias (SMQ) [Arrhythmia related investigations, signs and symptoms (SMQ); Cardiac arrhythmia terms (incl bradyarrhythmias and tachyarrhythmias) (SMQ)]; Cardiac failure (SMQ); Cardiomyopathy (SMQ); Ischaemic heart disease (SMQ)[ Myocardial infarction (SMQ)]; Shock (SMQ)[ Shock-associated circulatory or cardiac conditions (excl torsade de pointes) (SMQ)]; Torsade de pointes/QT prolongation (SMQ); Please see Appendix 3 |
| Increased Bilirubin | MedDRA PTs | Bilirubin conjugated abnormal Bilirubin conjugated increased Bilirubin excretion disorder Bilirubinuria Blood bilirubin abnormal Blood bilirubin increased Blood bilirubin unconjugated increased Hyperbilirubinaemia Icterus index increased Jaundice Jaundice cholestatic Jaundice extrahepatic obstructive Jaundice hepatocellular Ocular icterus Urine bilirubin increased Yellow skin |
| Events of clinical interest | | |
| Rash (all type) | MedDRA<br>HLTs, PTs | Erythemas - HLT Papulosquamous conditions - HLT Rashes, eruptions and exanthems NEC - HLT PT: Photodermatosis |

| | | Photosensitivity reaction |
|---|---|---|
| | | Polymorphic light eruption |
| | | Solar dermatitis |
| | | Sunburn |
| | SMQ | SMQ-Severe cutaneous adverse reaction: All |
| | | narrow terms and selected broad terms (refer |
| | | APPENDIX 2B below) |
| Pruritus | MedDRA HLT | Pruritus NEC |
| | | Photodermatosis |
| | | Photosensitivity reaction |
| Photosensitivity conditions | MedDRA PTs | Polymorphic light eruption |
| | | Solar dermatitis |
| | | Sunburn |

### 11.4.2 RASH – SMQ19.1

SMQ 19.1: "Severe cutaneous adverse reaction": all narrow and selected broad terms

| SCOPE | Preferred Term |
|--------|-------------------------------------------------------|
| NARROW | CUTANEOUS VASCULITIS |
| NARROW | DERMATITIS BULLOUS |
| NARROW | DERMATITIS EXFOLIATIVE |
| NARROW | DERMATITIS EXFOLIATIVE GENERALISED |
| NARROW | ERYTHEMA MULTIFORME |
| NARROW | OCULOMUCOCUTANEOUS SYNDROME |
| NARROW | SKIN NECROSIS |
| NARROW | STEVENS-JOHNSON SYNDROME |
| NARROW | TOXIC EPIDERMAL NECROLYSIS |
| NARROW | ACUTE GENERALISED EXANTHEMATOUS PUSTULOSIS |
| NARROW | TOXIC SKIN ERUPTION |
| NARROW | EPIDERMAL NECROSIS |
| NARROW | EXFOLIATIVE RASH |
| NARROW | DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS |
| BROAD | BLISTER |
| BROAD | BULLOUS IMPETIGO |
| BROAD | DRUG ERUPTION |
| BROAD | EPIDERMOLYSIS BULLOSA |
| BROAD | MUCOCUTANEOUS ULCERATION |
| BROAD | NIKOLSKY'S SIGN |
| BROAD | PEMPHIGOID |
| BROAD | PEMPHIGUS |
| BROAD | SKIN EROSION |
| BROAD | SKIN EXFOLIATION |
| BROAD | EPIDERMOLYSIS |
| BROAD | ACQUIRED EPIDERMOLYSIS BULLOSA |

## 11.4.3 CARDIAC EVENTS - SMQ19.1

| | Narrow/Broad | PT Term |
|---|---|---|
| | ythmias (SMQ) | |
| Arrhythi | mia related investig | ations, signs and symptoms (SMQ) |
| | Narrow | Chronotropic incompetence |
| | Narrow | Electrocardiogram repolarisation abnormality |
| | Narrow | Electrocardiogram RR interval prolonged |
| | Narrow | Electrocardiogram U-wave abnormality |
| | Narrow | Sudden cardiac death |
| | Broad | Bezold-Jarisch reflex |
| | Broad | Bradycardia |
| | Broad | Cardiac arrest |
| | Broad | Cardiac death |
| | Broad | Cardiac telemetry abnormal |
| | Broad | Cardio-respiratory arrest |
| | Broad | Central bradycardia |
| | Broad | Electrocardiogram abnormal |
| | Broad | Electrocardiogram ambulatory abnormal |
| | Broad | Electrocardiogram change |
| | Broad | Heart rate abnormal |
| | Broad | Heart rate decreased |
| | Broad | Heart rate increased |
| | Broad | Loss of consciousness |
| | Broad | Palpitations |
| | Broad | Rebound tachycardia |
| | Broad | Sudden death |
| | Broad | Syncope |
| | Broad | Tachycardia |
| | Broad | Tachycardia paroxysmal |
| Cardiac | arrhythmia terms ( | incl bradyarrhythmias and tachyarrhythmia |
| (SMQ) | | |
| | | conduction defects and disorders of sinus no |
| | ion) (SMQ) | |
| F | Bradyarrhythmia te | erms, nonspecific (SMQ) |
| | Narrow | Bradyarrhythmia |
| | Narrow | Ventricular asystole |
| | Conduction defects | |
| | Narrow | Accessory cardiac pathway |
| | Narrow | Adams-Stokes syndrome |
| | Narrow | Agonal rhythm |

| | Narrow | Atrial conduction time prolongation |
|----|---------------------|----------------------------------------------|
| | Narrow | Atrioventricular block |
| | Narrow | Atrioventricular block complete |
| | Narrow | Atrioventricular block first degree |
| | Narrow | Atrioventricular block second degree |
| | Narrow | Atrioventricular conduction time shortened |
| | Narrow | Atrioventricular dissociation |
| | Narrow | Bifascicular block |
| | Narrow | Brugada syndrome |
| | Narrow | Bundle branch block |
| | Narrow | Bundle branch block bilateral |
| | Narrow | Bundle branch block left |
| | Narrow | Bundle branch block right |
| | Narrow | Conduction disorder |
| | Narrow | Defect conduction intraventricular |
| | Narrow | Electrocardiogram delta waves abnormal |
| | Narrow | Electrocardiogram PQ interval prolonged |
| | Narrow | Electrocardiogram PQ interval shortened |
| | Narrow | Electrocardiogram PR prolongation |
| | Narrow | Electrocardiogram PR shortened |
| | Narrow | Electrocardiogram QRS complex prolonged |
| | Narrow | Electrocardiogram QT prolonged |
| | Narrow | Electrocardiogram repolarisation abnormality |
| | Narrow | Lenegre's disease |
| | Narrow | Long QT syndrome |
| | Narrow | Paroxysmal atrioventricular block |
| | Narrow | Sinoatrial block |
| | Narrow | Trifascicular block |
| | Narrow | Ventricular dyssynchrony |
| | Narrow | Wolff-Parkinson-White syndrome |
| | Disorders of sinus | s node function (SMQ) |
| | Narrow | Nodal arrhythmia |
| | Narrow | Nodal rhythm |
| | Narrow | Sinus arrest |
| | Narrow | Sinus arrhythmia |
| | Narrow | Sinus bradycardia |
| | Narrow | Sinus node dysfunction |
| | Narrow | Wandering pacemaker |
| Ca | ardiac arrhythmia t | erms, nonspecific (SMQ) |
| | Narrow | Arrhythmia |
| | | • |

| | Narrow | Heart alternation |
|-----|--------------------|---------------------------------------|
| | Narrow | Heart rate irregular |
| | Narrow | Pacemaker generated arrhythmia |
| | Narrow | Pacemaker syndrome |
| | Narrow | Paroxysmal arrhythmia |
| | Narrow | Pulseless electrical activity |
| | Narrow | Reperfusion arrhythmia |
| | Narrow | Withdrawal arrhythmia |
| Tac | | cl supraventricular and ventricular |
| | hyarrhythmias) (SI | - |
| | • • • • • | tachyarrhythmias (SMQ) |
| | Narrow | Arrhythmia supraventricular |
| | Narrow | Atrial fibrillation |
| | Narrow | Atrial flutter |
| | Narrow | Atrial parasystole |
| | Narrow | Atrial tachycardia |
| | Narrow | Junctional ectopic tachycardia |
| | Narrow | Sinus tachycardia |
| | Narrow | Supraventricular extrasystoles |
| | Narrow | Supraventricular tachyarrhythmia |
| | Narrow | Supraventricular tachycardia |
| | Broad | ECG P wave inverted |
| | Broad | Electrocardiogram P wave abnormal |
| | Broad | Retrograde p-waves |
| | Tachyarrhythmia | terms, nonspecific (SMQ) |
| | Narrow | Anomalous atrioventricular excitation |
| | Narrow | Cardiac fibrillation |
| | Narrow | Cardiac flutter |
| | Narrow | Extrasystoles |
| | Narrow | Tachyarrhythmia |
| | | varrhythmias (SMQ) |
| | Narrow | Accelerated idioventricular rhythm |
| | Narrow | Cardiac fibrillation |
| | Narrow | Parasystole |
| | Narrow | Rhythm idioventricular |
| | Narrow | Torsade de pointes |
| | Narrow | Ventricular arrhythmia |
| | Narrow | Ventricular extrasystoles |
| | Narrow | Ventricular fibrillation |
| | Narrow | Ventricular flutter |

| | Narrow | Ventricular parasystole |
|------------|-------------|-----------------------------------------------|
| | Narrow | Ventricular pre-excitation |
| | Narrow | Ventricular tachyarrhythmia |
| | Narrow | Ventricular tachycardia |
| Cardiac fa | ilure (SMQ) | , |
| | Narrow | Acute left ventricular failure |
| | Narrow | Acute pulmonary oedema |
| | Narrow | Acute right ventricular failure |
| | Narrow | Cardiac asthma |
| | Narrow | Cardiac failure |
| | Narrow | Cardiac failure acute |
| | Narrow | Cardiac failure chronic |
| | Narrow | Cardiac failure congestive |
| | Narrow | Cardiac failure high output |
| | Narrow | Cardiogenic shock |
| | Narrow | Cardiopulmonary failure |
| | Narrow | Cardiorenal syndrome |
| | Narrow | Chronic left ventricular failure |
| | Narrow | Chronic right ventricular failure |
| | Narrow | Cor pulmonale |
| | Narrow | Cor pulmonale acute |
| | Narrow | Cor pulmonale chronic |
| | Narrow | Ejection fraction decreased |
| | Narrow | Hepatic congestion |
| | Narrow | Hepatojugular reflux |
| | Narrow | Left ventricular failure |
| | Narrow | Low cardiac output syndrome |
| | Narrow | Neonatal cardiac failure |
| | Narrow | Obstructive shock |
| | Narrow | Pulmonary oedema |
| | Narrow | Pulmonary oedema neonatal |
| | Narrow | Radiation associated cardiac failure |
| | Narrow | Right ventricular ejection fraction decreased |
| | Narrow | Right ventricular failure |
| | Narrow | Ventricular failure |
| | Broad | Artificial heart implant |
| | Broad | Atrial natriuretic peptide abnormal |
| | Broad | Atrial natriuretic peptide increased |
| | Broad | Bendopnoea |
| | Broad | Brain natriuretic peptide abnormal |

| Broad | Brain natriuretic peptide increased |
|-------|-------------------------------------------------|
| Broad | |
| Broad | |
| Broad | |
| Broad | 1 |
| Broad | |
| Broad | |
| Broad | |
| Broad | 8 8 |
| Broad | |
| Broad | 1 2 |
| Broad | |
| Broad | Central venous pressure increased |
| Broad | · |
| Broad | Dilatation ventricular |
| Broad | Dyspnoea paroxysmal nocturnal |
| Broad | Heart transplant |
| Broad | Hepatic vein dilatation |
| Broad | Jugular vein distension |
| Broad | Left ventricular dilatation |
| Broad | Left ventricular dysfunction |
| Broad | Left ventricular enlargement |
| Broad | Lower respiratory tract congestion |
| Broad | Myocardial depression |
| Broad | Nocturnal dyspnoea |
| | N-terminal prohormone brain natriuretic peptide |
| Broad | abnormal |
| | N-terminal prohormone brain natriuretic peptide |
| Broad | increased |
| Broad | Oedema |
| Broad | Oedema due to cardiac disease |
| Broad | Oedema neonatal |
| Broad | Oedema peripheral |
| Broad | Orthopnoea |
| Broad | Peripheral oedema neonatal |
| Broad | |
| Broad | Post cardiac arrest syndrome |
| Broad | Prohormone brain natriuretic peptide abnormal |
| Broad | |
| Broad | * * |

| | Broad | Right ventricular dilatation |
|---|---|---|
| | Broad | Right ventricular dysfunction |
| | Broad | Right ventricular dystanction Right ventricular enlargement |
| | Broad | Scan myocardial perfusion abnormal |
| | Broad | Stroke volume decreased |
| | Broad | |
| | Broad | Surgical ventricular restoration |
| | Broad | Systolic dysfunction |
| | | Venous pressure increased |
| | Broad | Venous pressure jugular abnormal |
| | Broad | Venous pressure jugular increased |
| | Broad | Ventricular assist device insertion |
| | Broad | Ventricular dysfunction |
| | Broad | Ventricular dyssynchrony |
| Cardiomyo | pathy (SMQ) | |
| | Narrow | Atrial septal defect acquired |
| | Narrow | Biopsy heart abnormal |
| | Narrow | Cardiac amyloidosis |
| | Narrow | Cardiac hypertrophy |
| | Narrow | Cardiac sarcoidosis |
| | Narrow | Cardiac septal hypertrophy |
| | Narrow | Cardiac siderosis |
| | Narrow | Cardiomyopathy |
| | Narrow | Cardiomyopathy acute |
| | Narrow | Cardiomyopathy alcoholic |
| | Narrow | Cardiomyopathy neonatal |
| | Narrow | Cardiotoxicity |
| | Narrow | Congestive cardiomyopathy |
| | Narrow | Cytotoxic cardiomyopathy |
| | Narrow | Diabetic cardiomyopathy |
| | Narrow | Ejection fraction abnormal |
| | Narrow | Ejection fraction decreased |
| | Narrow | Eosinophilic myocarditis |
| | Narrow | HIV cardiomyopathy |
| | Narrow | Hypertensive cardiomyopathy |
| | Narrow | Hypertrophic cardiomyopathy |
| | Narrow | Ischaemic cardiomyopathy |
| | Narrow | Metabolic cardiomyopathy |
| | Narrow | Myocardial calcification |
| | Narrow | Myocardial fibrosis |
| | Narrow | Myocardial haemorrhage |
| | 11411011 | 1.1,000itatui itaoinoititugo |

| Narrow | Non-obstructive cardiomyopathy |
|--------|-----------------------------------------------|
| Narrow | Peripartum cardiomyopathy |
| Narrow | Pulmonary arterial wedge pressure increased |
| Narrow | Restrictive cardiomyopathy |
| Narrow | Right ventricular ejection fraction decreased |
| Narrow | Stress cardiomyopathy |
| Narrow | Tachycardia induced cardiomyopathy |
| Narrow | Thyrotoxic cardiomyopathy |
| Narrow | Ventricular septal defect acquired |
| Narrow | Viral cardiomyopathy |
| Broad | Abnormal precordial movement |
| Broad | Acquired cardiac septal defect |
| Broad | Acute left ventricular failure |
| Broad | Alcohol septal ablation |
| Broad | Allergic myocarditis |
| Broad | Arrhythmia |
| Broad | Arrhythmia supraventricular |
| Broad | Artificial heart implant |
| Broad | Ascites |
| Broad | Atrial hypertrophy |
| Broad | Atrial pressure increased |
| Broad | Autoimmune myocarditis |
| Broad | Bendopnoea Bendopnoea |
| Broad | Blood pressure diastolic abnormal |
| Broad | Blood pressure diastolic decreased |
| Broad | Blood pressure diastolic increased |
| Broad | Blood pressure fluctuation |
| Broad | Blood pressure inadequately controlled |
| Broad | Blood pressure systolic abnormal |
| Broad | Blood pressure systolic decreased |
| Broad | Blood pressure systolic increased |
| Broad | Cardiac aneurysm |
| Broad | Cardiac arrest |
| Broad | Cardiac contractility modulation therapy |
| Broad | Cardiac electrophysiologic study abnormal |
| Broad | Cardiac failure |
| Broad | Cardiac failure acute |
| Broad | Cardiac failure chronic |
| Broad | Cardiac failure congestive |
| Broad | Cardiac function test abnormal |
| Dioud | Cardiae Iditeriori teot aoriorinar |

| | Broad | Cardiac imaging procedure abnormal |
|---|---|---|
| | Broad | Cardiac index abnormal |
| | Broad | Cardiac index decreased |
| | Broad | Cardiac index increased |
| | Broad | Cardiac monitoring abnormal |
| | Broad | Cardiac operation |
| | Broad | Cardiac output decreased |
| | Broad | Cardiac pseudoaneurysm |
| | Broad | Cardiac resynchronisation therapy |
| | Broad | Cardiac ventricular scarring |
| | Broad | Cardiac ventriculogram abnormal |
| | Broad | Cardiac ventriculogram left abnormal |
| | Broad | Cardiac ventriculogram right abnormal |
| <del> </del> | Broad | Cardiomegaly |
| | Broad | Cardiothoracic ratio increased |
| | Broad | Cardiovascular disorder |
| | Broad | Cardiovascular function test abnormal |
| | Broad | Chest pain |
| | Broad | Chest X-ray abnormal |
| | Broad | Computerised tomogram thorax abnormal |
| | Broad | Coxsackie carditis |
| | Broad | Coxsackie myocarditis |
| | Broad | Cytomegalovirus myocarditis |
| | Broad | Decreased ventricular preload |
| | Broad | Diastolic dysfunction |
| | Broad | Dilatation atrial |
| | Broad | Dilatation ventricular |
| | Broad | Directional Doppler flow tests abnormal |
| | Broad | Dyspnoea |
| | Broad | ECG signs of ventricular hypertrophy |
| | Broad | Echocardiogram abnormal |
| | Broad | Electrocardiogram abnormal |
| | Broad | Electrocardiogram change |
| | Broad | Endocardial fibroelastosis |
| | Broad | External counterpulsation |
| | Broad | Gonococcal heart disease |
| <del> </del> | Broad | Heart and lung transplant |
| <del> </del> | Broad | Heart transplant |
| | Broad | Hepatomegaly |
| | Broad | Hyperdynamic left ventricle |
| | Diouu | 11) potaj namio toti vontitoto |

| Broad | Increased ventricular preload |
|-------|---------------------------------------------|
| Broad | Irregular breathing |
| Broad | Labile blood pressure |
| Broad | Left atrial dilatation |
| Broad | Left atrial enlargement |
| Broad | Left ventricular dilatation |
| - 1 | Left ventricular end-diastolic pressure |
| Broad | decreased |
| Broad | Left ventricular enlargement |
| Broad | Left ventricular failure |
| Broad | Left ventricular heave |
| Broad | Lupus myocarditis |
| Broad | Lyme carditis |
| Broad | Malarial myocarditis |
| Broad | Mental status changes |
| Broad | Multiple gated acquisition scan abnormal |
| Broad | Myocardiac abscess |
| Broad | Myocardial necrosis marker increased |
| Broad | Myocarditis |
| Broad | Myocarditis bacterial |
| Broad | Myocarditis helminthic |
| Broad | Myocarditis infectious |
| Broad | Myocarditis meningococcal |
| Broad | Myocarditis mycotic |
| Broad | Myocarditis post infection |
| Broad | Myocarditis septic |
| Broad | Myocarditis syphilitic |
| Broad | Myocarditis toxoplasmal |
| Broad | Myoglobinaemia |
| Broad | Myoglobinuria |
| Broad | Nocturia |
| | Nuclear magnetic resonance imaging thoracic |
| Broad | abnormal |
| Broad | Oedema |
| Broad | Orthostatic hypotension |
| Broad | Palpitations |
| Broad | Papillary muscle disorder |
| Broad | Papillary muscle haemorrhage |
| Broad | Radiation myocarditis |
| Broad | Right atrial dilatation |
| Divau | ragin untai unatation |

| | Broad | Right atrial enlargement |
|---|---|---|
| | Broad | Right atrial pressure increased |
| | Broad | Right ventricle outflow tract obstruction |
| | Broad | Right ventricular dilatation |
| | Broad<br>Broad | Right ventricular enlargement |
| | | Right ventricular heave |
| | Broad | Right ventricular systolic pressure decreased |
| | Broad | Scan myocardial perfusion abnormal |
| | Broad | Sudden cardiac death |
| | Broad | Sudden death |
| | Broad | Surgical ventricular restoration |
| | Broad | Syncope |
| | Broad | Systolic anterior motion of mitral valve |
| | Broad | Systolic dysfunction |
| | Broad | Ultrasound Doppler abnormal |
| | Broad | Vascular resistance pulmonary increased |
| | Broad | Ventricular arrhythmia |
| | Broad | Ventricular assist device insertion |
| | Broad | Ventricular dysfunction |
| | Broad | Ventricular dyskinesia |
| | Broad | Ventricular dyssynchrony |
| | Broad | Ventricular hyperkinesia |
| | Broad | Ventricular hypertrophy |
| | Broad | Ventricular hypokinesia |
| | Broad | Ventricular remodelling |
| | Broad | Viral myocarditis |
| Ischaemic hea | rt disease (SMQ) | |
| Myocardi | al infarction (SMQ | ) |
| | Narrow | Acute coronary syndrome |
| | Narrow | Acute myocardial infarction |
| | Narrow | Angina unstable |
| | Narrow | Blood creatine phosphokinase MB abnormal |
| | Narrow | Blood creatine phosphokinase MB increased |
| | Narrow | Coronary artery embolism |
| | Narrow | Coronary artery occlusion |
| | Narrow | Coronary artery reocclusion |
| | Narrow | Coronary artery thrombosis |
| | Narrow | Coronary bypass thrombosis |
| | Narrow | Coronary vascular graft occlusion |
| | Narrow | Kounis syndrome |
| | 1 | <u> </u> |

| | Narrow | Myocardial infarction |
|---|---|---|
| | Narrow | Myocardial necrosis |
| <del>- - -</del> | Narrow | Myocardial reperfusion injury |
| | Narrow | Myocardial stunning |
| | Narrow | Papillary muscle infarction |
| | Narrow | Post procedural myocardial infarction |
| | Narrow | Postinfarction angina |
| | Narrow | Silent myocardial infarction |
| | Narrow | Troponin I increased |
| | Narrow | Troponin increased Troponin increased |
| | Narrow | Troponin T increased |
| | Broad | Blood creatine phosphokinase abnormal |
| | Broad | Blood creatine phosphokinase abnormal |
| | Broad | Cardiac ventricular scarring |
| | Broad | ECG electrically inactive area |
| | Broad | ECG electrically inactive area ECG signs of myocardial infarction |
| | Broad | Electrocardiogram Q wave abnormal |
| | Broad | Electrocardiogram ST segment abnormal |
| | Broad | Electrocardiogram ST segment abnormal Electrocardiogram ST segment elevation |
| | Broad | Electrocardiogram ST-T segment elevation |
| | Broad | Infarction |
| | Broad | Myocardial necrosis marker increased |
| | Broad | - |
| | | Scan myocardial perfusion abnormal |
| | Broad | Vascular graft occlusion |
| | Broad | Vascular stent occlusion |
| GL 1 (CMO) | Broad | Vascular stent thrombosis |
| | Narrow | Acute left ventricular failure |
| | Narrow | Adams-Stokes syndrome |
| | Narrow | Atrial parasystole |
| | Narrow | Cardiac arrest |
| | Narrow | Cardiac arrest neonatal |
| | Narrow | Cardiac death |
| | Narrow | Cardiac fibrillation |
| | Narrow | Cardiac flutter |
| | Narrow | Cardiogenic shock |
| | Narrow | Cardio-respiratory arrest |
| | Narrow | Cardio-respiratory arrest neonatal |

| | Narrow | Cardiovascular insufficiency |
|---------------|-------------------|----------------------------------------|
| | Narrow | Circulatory collapse |
| | Narrow | Obstructive shock |
| | Narrow | Pulse absent |
| | - 1.00-2-0-11 | |
| | Narrow | Pulseless electrical activity |
| | Narrow | Shock |
| | Narrow | Shock symptom |
| | Narrow | Sudden cardiac death |
| | Narrow | Ventricular asystole |
| | Narrow | Ventricular fibrillation |
| | Narrow | Ventricular flutter |
| | Narrow | Ventricular parasystole |
| | Broad | Acute kidney injury |
| | Broad | Acute prerenal failure |
| | Broad | Acute respiratory failure |
| | Broad | Anuria |
| | Broad | Blood pressure immeasurable |
| | Broad | Cerebral hypoperfusion |
| | Broad | Grey syndrome neonatal |
| | Broad | Hepatic congestion |
| | Broad | Hepatojugular reflux |
| | Broad | Hepatorenal failure |
| | Broad | Hypoperfusion |
| | Broad | Jugular vein distension |
| | Broad | Myocardial depression |
| | Broad | Neonatal anuria |
| | Broad | Neonatal multi-organ failure |
| | Broad | Neonatal respiratory failure |
| | Broad | Organ failure |
| | Broad | Prerenal failure |
| | Broad | Propofol infusion syndrome |
| | Broad | Renal failure |
| | Broad | Renal failure neonatal |
| | Broad | Respiratory failure |
| Torsade de po | intes/QT prolonga | |
| | Narrow | Electrocardiogram QT interval abnormal |
| | Narrow | Electrocardiogram QT prolonged |
| | Narrow | Long QT syndrome |
| | Narrow | Long QT syndrome congenital |
| | Narrow | Torsade de pointes |
| | L | * |

| Narrow | Ventricular tachycardia |
|--------|----------------------------------------------|
| Broad | Cardiac arrest |
| Broad | Cardiac death |
| Broad | Cardiac fibrillation |
| Broad | Cardio-respiratory arrest |
| Broad | Electrocardiogram repolarisation abnormality |
| Broad | Electrocardiogram U-wave abnormality |
| Broad | Loss of consciousness |
| Broad | Sudden cardiac death |
| Broad | Sudden death |
| Broad | Syncope |
| Broad | Ventricular arrhythmia |
| Broad | Ventricular fibrillation |
| Broad | Ventricular flutter |
| Broad | Ventricular tachyarrhythmia |